

# **Groupe Axonal-Biostatem**

Parc d'activités Via Domitia 205, avenue des Gardians 34160 CASTRIES - FRANCE 2: 33 (0) 4 67 04 87 54

**≞**: 33 (0) 4 67 04 87 71

E-mail: contact@biostatem.com



#### **Sponsor**

Laboratoires THÉA
Research and Development Department
12, rue Louis Blériot
63017 Clermont-Ferrand Cedex 2, France



# STATISTICAL ANALYSIS PLAN

Comparison of the performance and safety of T2259 versus Vismed® Multi in dry eye patients with superficial keratitis.

**Investigation No. LT2259-001** 

Ref Axonal-Biostatem: E876

Type of study: Investigation (Medical device)

Statistician:

Version number: No. 1.2

Date of issue: 01JUL2021

Type of report: Final

# **HISTORY OF THE VERSIONS**

| Version | Concerned parts | Date | Nature <sup>(*)</sup> | Reasons of change |
|---|---|---|---|---|
| Draft 0.1 | All | 03SEP2020 | С | |
| Draft 0.2 | All | 27JAN2021 | М | Review of the sponsor |
| Draft 0.3 | All | 28APR2021 | М | Review of the sponsor |
| Draft 0.4 | All | 10JUN2021 | M | Review of the sponsor |
| Final 1.0 | All | 16JUN2021 | M | Review of the sponsor |
| Final 1.1 | All | 29JUN2021 | М | Review of MW and biostatistician |
| Final 1.2 | All | 01JUL2021 | М | Review of sponsor for consistency |

 $<sup>^{(*)}</sup>$  C: Creation, M: Modification, A: Addition, D: Delete

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

# **SIGNATURE FORM**

| Author of the Statistical Analysis Plan: | (statistician, Axonal-Biostatem) |
|------------------------------------------|----------------------------------|
| Date: | |
| Signature: | |

Proofreading and validation by Axonal-Biostatem:



# **TABLES OF CONTENTS**

| 1 | STU | DY OBJECTIVES | 8 |
|---|---|---|---|
| | 1.1 | Primary objective | 8 |
| | 1.2 | Secondary objective | 8 |
| 2 | STU | DY DESIGN | 8 |
| | 2.1 | Overview | 8 |
| | 2.2 | Study population | <u>S</u> |
| | 2.2.1 | Inclusion criteria | <u>S</u> |
| | 2.2.2 | Exclusion criteria | <u>S</u> |
| | 2.3 | Investigational Medical Devices | 11 |
| | 2.4 | Randomisation | |
| | 2.5 | Study schedule | 13 |
| 3 | STUI | DY OUTCOME VARIABLES | 16 |
| | 3.1 | Performance criteria | 16 |
| | 3.1.1 | Primary performance endpoint | 16 |
| | 3.1.2 | | |
| | 3.2 | Safety assessments | 16 |
| | 3.3 | Derived variables | 17 |
| 4 | SEQI | JENCE OF PLANNED ANALYSES | 27 |
| | 4.1 | Interim analyses | 27 |
| | 4.2 | Final analyses and reporting | 27 |
| | 4.3 | Changes to statistical information in the clinical trial protocol | |
| 5 | STAT | ISTICAL METHODOLOGY | |
| | 5.1 | Detailed power and sample size | 28 |
| | 5.2 | Generalities for statistical analyses | 28 |
| | 5.3 | Multiple Imputations for Handling of Dropouts or Missing data | 30 |
| | 5.4 | Adjustments for Covariates | 31 |
| | 5.5 | Multicentre | 31 |
| 6 | STAT | ISTICAL ANALYSES | 31 |
| | 6.1 | Study Populations | 31 |
| | 6.1.1 | Protocol Deviations | 31 |
| | 6.1.2 | Analysis Populations | 32 |
| | 6.2 | Disposition of Patients | 33 |
| | 6.3 | Demographic and Baseline Characteristics | 35 |
| | 6.4 | Subgroup analysis | 35 |
| | 6.5 | Previous, Concomitant and Post-Study Medications | 36 |
| | 6.6 | Treatment exposure and compliance | 36 |
| | 6.7 | Performance analyses | 37 |
| | 6.7.1 | Primary Performance Endpoint | 37 |
| | 6.7.2 | Secondary Performance Endpoints | 39 |
| | 6.8 | Safety Analysis | 41 |
| | 6.8.1 | Safety endpoints | 41 |
| | 6.8.2 | Adverse events | 42 |
| | 6.8.3 | Device deficiencies | 44 |
| 7 | REPO | DRTING CONVENTIONS | 44 |
| | 7.1 | Software used | 44 |

| Statistical analysis plan | | 01JUL2021 |
|---------------------------|------------------------|---------------|
| E876 | | SAP Final 1.2 |
| 7.2 | General considerations | 44 |

| | 7.2 | General considerations | . 44 |
|----|-------|----------------------------------------------------------|------|
| | 7.3 | Statistical summary conventions | . 44 |
| | 7.4 | Examples of tables, listings and figures | . 44 |
| | 7.4.2 | 1 Quantitative variables | . 44 |
| | 7.4.2 | 2 Qualitative variables | . 45 |
| | 7.4.3 | B Protocol deviations | . 47 |
| | 7.4.4 | 4 Adverse Events | . 47 |
| 8 | TAB | LES, LISTING AND FIGURES | . 49 |
| | 8.1 | Planned tables | . 49 |
| | 8.2 | Planned listings | . 56 |
| | 8.3 | Planned figures | . 57 |
| 9 | REFE | ERENCES | . 58 |
| 1( | ) APP | ENDICES | . 59 |
| | 10.1 | Appendix 1: Level of validation for analyses programming | . 59 |

# LIST OF ABBREVIATIONS

**95% CI** 95% Confidence Interval

AE Adverse Events

ADE Adverse Device Effect

ATC Anatomical Therapeutic Chemical Classification

**ANCOVA** Analysis of Covariance

AUF Arbitrary Units of Fluorescence
BCVA Far Best-corrected visual acuity

**BR** Blind Review

CI Confidence interval

COVID Corona Virus Disease
CSR Clinical Study Report

**D1, D8, D35, D84** Day 1/8/35/84

DEQ-5
 e-CRF
 Electronic Case Report Form
 CRO
 Contract Research Organisation

**FAS** Full Analysis Set

FPFV First Patient First Visit
FPLV First Patient Last Visit

HLA-DR Human Leukocyte Antigen – antigen D Related ICH International Conference of Harmonisation

IMD Investigational Medical Device
IWRS Interactive Response System

**LOCF** Last Observation Carried Forward

LPFV Last Patient First Visit
LPLV Last Patient Last Visit

LE Least Square MD Medical Device

MedDRA Medical Dictionary for Regulatory Activities

Min.; Max. Minimum; Maximum

MMRM Mixed Model for Repeated Measures

OSI Optical Scattering Index

OSDI Ocular Surface Disease Index
OQAS Optical Quality Analysing System

PP Per Protocol
PT Preferred Term

Q1; Q3 First Quartile; Third Quartile
SADE Serious Adverse Device Effect

SAE Serious Adverse Event

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

| SAF | Safety (population) |
|------|-----------------------------------|
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TBUT | Tear Break-up Time |
| TEAE | Treatment emergent adverse events |
| WHO | World Health Organisation |

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

The Statistical analysis Plan (SAP) aims to describe the statistical analyses that will be performed for the study LT2259-001, based on the study protocol (Version 3.0 – 3 January 2020) and the e-Case Report Form (e-CRF) (Version MSC003, dated on 06 APR 2020), in accordance with ICH Guidelines and the general statistical principles.

This document is written by the AXONAL-BIOSTATEM statistician and reviewed and approved by the Sponsor of the Investigation (Laboratoires Théa) before the database lock.

#### 1 STUDY OBJECTIVES

## 1.1 Primary objective

The primary objective of this study is to demonstrate the non-inferiority of T2259 versus Vismed® Multi in terms of performance.

Non-inferiority will be tested by calculating the bilateral 95% CI of the difference between groups (T2259 – Vismed® Multi) of the change from baseline of total ocular staining according to Oxford 0-15 grading scheme on Day 35. If the upper bound is no higher than 2 points, it will be concluded that the null hypothesis can be rejected and that the performance of T2259 is non-inferior to that of Vismed® Multi.

The non-inferiority analysis will be provided primarily in the PP population and confirmed in the FAS population.

# 1.2 Secondary objective

The secondary objective of the investigation is to evaluate the safety and the performance of T2259 versus Vismed® Multi.

# 2 STUDY DESIGN

#### 2.1 Overview

Day 84 (± 7)

This is a multicentre, randomised study, investigator-masked, 2 parallel groups (T2259 versus Vismed® Multi) of 38 evaluable patients each.

The patients were randomised after a run-in-period of 7 to 10 days with preservative free artificial tears (Hydrabak®, one drop in each eye 3 to 6 times daily). Then, they were treated with either T2259 or the reference product (Vismed® Multi) for 84 days (± 7 days).

Investigation visits were performed as following:

Final visit (Visit 5)

| Day 1-10/Day 1-7 | Selection visit (Visit 1) |
|---|---|
| Day 1 | Randomisation/ Inclusion visit (Visit 2) |
| Day 8 (± 1) | Visit 3 Optional Visit (if the investigator and/or the patient thinks it |
| | is necessary) |
| Day 35 (± 3) | Visit 4 |


The Visits V2, V3, V4 and V5 should have been performed at the same hour (±4 hours).

#### Reclassification of visits:

All "premature withdrawal" visits will be reclassified as decided in BR Meeting. Number of days between premature withdrawal visits and randomisation visit will be calculated and depending of this number of days, visits will be reclassified to the nearest planned non-missing visit.

# 2.2 Study population

## 2.2.1 Inclusion criteria

At selection visit (Day 1-10/Day 1-7):

- Informed consent signed and dated.
- Male or female aged ≥ 18 years old.
- Known Dry Eye Syndrome requiring artificial tears within the last 3 months prior to study selection.

## At randomisation visit (Day 1):

- Patient having used only unpreserved artificial tears (Hydrabak®) as ocular medication during the run-in period (from Day 1-10/Day 1 -7 to Day 1).
- No ocular instillation at least 6 hours prior to the randomisation visit (Day 1).
- Diagnosis of moderate to severe dry eye syndrome defined by OSDI Score ≥ 23.
- Patients having at least one Eligible Eye, defined by both following conditions:
  - $\circ$  Total ocular staining (corneal and conjunctival) with Oxford 0- 15 grading scheme ≥ 4 and ≤ 9.

## AND

- At least one of the following objective signs:
  - Schirmer test ≥ 3 mm/5 min and ≤ 9 mm/5 min Or
  - TBUT: sum of 3 measurements ≤ 30 seconds.

#### 2.2.2 <u>Exclusion criteria</u>

# Ophthalmic Exclusion Criteria in AT LEAST ONE EYE:

- Far best-corrected visual acuity ≤ 2/10.
- Severe blepharitis (grade 3 / 0-3 scale).
- Ocular rosacea.
- Severe Dry Eye associated to:
  - Eyelid malposition,
  - Corneal dystrophy,
  - Ocular neoplasia,

- Filamentous keratitis,
- Corneal neovascularisation,
- Orbital radiotherapy.
- History of ocular trauma, ocular infection or ocular inflammation within the last 3 months.
- History of ocular allergy.
- History of uveitis.
- History of inflammatory corneal ulcer within the last 12 months.
- Glaucoma, ocular hypertension requiring glaucoma treatment.

# Systemic/Non-Ophthalmic Exclusion Criteria:

- Known or suspected hypersensitivity to one of the components of the Investigational Device or auxiliary products.
- History of active relevant systemic condition incompatible with the study or likely to interfere with the study results or the patient safety according to investigator judgment.
- Allergic rhinitis active or susceptible to reactivate during the study.
- Any other medical or surgical history, disorder or disease susceptible to require or to modify systemic medication during the study (systemic medication having to be stable within the three months before selection).

# <u>Specific Exclusion Criteria Regarding Childbearing Potential Women:</u>

- Pregnancy or breastfeeding.
- Childbearing potential woman who is not using a reliable method of contraception (oral contraceptive, intra-uterine device, subcutaneous contraceptive implant, vaginal ring, patch) and is not surgically sterilised.

#### Exclusion Criteria Related to General Conditions

- Inability of patient to understand the study procedures or to give informed consent.
- Non-compliant patient (e.g., not willing to attend a visit or completing the self-questionnaire; way of life interfering with compliance).
- Participation in this investigation at the same time as another clinical investigation.
- Participation in this investigation during the exclusion period of another clinical study.
- Patient previously randomized in this study.
- Patient being institutionalized because of legal or regulatory order, inmate of psychiatric wards, prison or state institutions, or employee of the study sites or of the sponsor's company.
- Patient not covered by the government health care scheme of the country in which he/she is living.

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

- Patient under guardianship/ward of court

Exclusion criteria related to previous and concomitant treatments (medications/non-medicinal therapies/procedures)

- Patient with previous, current prohibited listed treatment (or prohibited modification of treatment regimen).

The prohibited treatments (or prohibited modifications of treatment regimen) and their periods of use prohibition are listed in the following table:

| CONCOMITANT MEDICATIONS/NON-MEDICINAL TREATMENTS NOT ALLOWED BEFORE AND DURING THE INVESTIGATION | | | | | | |
|---|---|---|---|---|---|---|
| Before the selection visit (Before Day 1-10/Day 1-7) | | | Run-in period (From<br>Day 1-10/Day 1-7 to<br>Day 1) | After<br>randomisation<br>(Day 1 to Day<br>84) | | |
| 12 months | 6 months | 3 months | 1 month | 1 week | Run-in period | Treatment period |
| Corneal surgery, | | | | | | |
| Intraocular injections | | | | | | |
| | | | | 250 | ral)<br>imus, pimecrolimus | |
| | Any change in systemic medication already ongoing before selection visit | | | | | |
| | | | Semi-per | manent o | r temporary punctal plugs | |
| | | | | Contact l | enses | |
| | Any ocular medication other than Hydrabak® | | | | | |
| | | | | | | Any ocular medication including artificial tears other than authorized medical devices |

# 2.3 Investigational Medical Devices

T2259

Formulation: Trehalose, 6%; Sodium Hyaluronate, 0.2%

Route of administration: Eye drops

Daily dose regimen: One drop in each eye 2 to 4 times daily

Vismed® Multi


Formulation: Sodium Hyaluronate, 0.18%

**Route of administration:** Eye drops

Daily dose regimen: One drop in each eye 2 to 4 times daily

#### 2.4 Randomisation

A patient who had given his/her written informed consent and who was included in the study was assigned a specific treatment number.

Random allocation of patients in the T2259 group or Vismed® Multi group assure that all patient's known and unknown characteristics are similar and balanced between groups at the beginning of the study, avoiding the selection bias.

The randomisation code list stratified by site was generated by the CRO in charge of the statistics (AXONAL-BIOSTATEM / independent statistician). Patients were randomised on a 1:1 basis to T2259 or comparator product respectively. The Investigational Medical Device (IMD) was allocated to the patients according to randomisation using an interactive response system (IWRS).

Randomisation occurred at the randomisation visit (Day 1; Visit 2) after all screening procedures had been performed and eligibility for the study confirmed. The patient who met the eligibility criteria was randomly assigned to treatment and associated to a randomisation number.

The treatment number should be recorded in patient's source documents and in the e-CRF.

During the visit 4 (Day 35), this investigator allocated the same treatment number than he did at the randomisation visit.

The treatment number must be recorded in the patient's source document and the e-CRF.

# 2.5 Study schedule

**Table 1: Study Schedule** 

| STUDY PROCEDURE | Visit #1<br>Selection visit<br>D1-10/D1-7 | Run-in<br>period | vi | t #2<br>nisation<br>sit | Visi<br>D8 (<br>Optiona | | | t #4<br>(± 3) | Visit<br>Final<br>D84 (<br>O<br>Prema<br>withdr | Visit<br>± 7)<br>r<br>ature |
|---|---|---|---|---|---|---|---|---|---|---|
| | First<br>ophthalmologist<br>investigator | | First ophthalmologist<br>investigator | Second investigator | First ophthalmologist<br>investigator | Second investigator | First ophthalmologist<br>investigator | Second investigator | First ophthalmologist<br>investigator | Second investigator |
| Informed consent | х | bak | ophthalmol<br>investigator | nve | halr | uve | ophthalmol | nve | ophthalmol | uve. |
| Demography | х | /dra | pht | i B | pht | nd i | pht | nd i | pht | i Bi |
| Ocular medical and surgical history | х | S H | rsto | 9 | rsto | eco | rsto | 960 | rsto | 9 |
| Systemic medical and surgical<br>history | х | ial tear | E | 0, | <u> </u> | , s, | Œ | 0, | Œ | , , |
| Previous and concomitant<br>ocular/non ocular treatments | х | Preservative free artificial tears Hydrabak® | х | | х | | х | | х | |
| History of Dry Eye | х | free | | | | | | | | |
| DEQ-5 | х | ive | | | | | х | | Х | |
| OSDI score | | ıvat | х | | х | | Х | | х | |
| Ocular symptoms | х | rese | х | | х | | х | | х | |
| Ocular symptoms upon instillation <sup>(2)</sup> | | Ā | | | | х | | X | | х |
| Far best-corrected visual acuity | х | | | | | | х | | х | |
| Conjunctival hyperaemia<br>(McMonnies photographic scale) | x | | х | | х | | х | | х | |

| Slit lamp examination | х | х | | х | | Х | | х | |
|---|---|---|---|---|---|---|---|---|---|
| TBUT | х | Х | | х | | х | | х | |
| Oxford 0-15 grading scheme<br>(corneal staining by<br>fluorescein, temporal and<br>nasal staining by lissamine) | х | х | | х | | х | | х | |
| Van Bijsterveld score<br>(lissamine green<br>staining)/optional<br>examination <sup>(7)</sup> | х | х | | х | | х | | х | |
| Schirmer test (without anaesthesia) | | х | | х | | х | | х | |
| Verification of inclusion/exclusion criteria | х | х | | | | | | | |
| Tolerance assessment by the investigator | | | | | | х | | х | |
| Tolerance assessment by the patient | | | | | | х | | х | |
| Performance assessment by the investigator | | | | | | х | | х | |
| Urinary pregnancy test (2) | х | | | | | х | | х | |
| Adverse events | | х | | х | х | х | х | х | х |
| Dispensation of the run-in treatment | х | | | | | | | | |
| Run-in treatment compliance | | х | | | | | | | |
| Dispensation of the IMD (3) | | | х | | ! | | х | | |
| IMD compliance (3) | | | | | | | х | | х |
| Evaluation of Optical Scattering<br>Index (OSI) using double pass<br>aberrometry <sup>(4)</sup> | | х | | | | х | | х | |

| Impression cytology (HLA-DR) Only | > | v |
|--------------------------------------|---|---|
| for patients with severe Dry Eye (5) | ^ | ^ |

- (1) No instillation of preservative free artificial tears (Hydrabak®) at least 6 hours before the randomisation visit.
- (2) Urinary pregnancy test to be done for childbearing potential women.
- (3) By the second investigator (or the designated site team member) responsible for dispensing, explications of dosing regimen,
- (4) The parameters will be measured only in investigator sites equipped with Optical Quality Analysing System (OQAS)
- (5) Severe Dry Eye will be defined based on the following criteria: OSDI≥33 and/or Corneal Fluorescein Staining ≥ 3 at the baseline visit (Day 1).
- (6) This visit can be performed if the investigator and/or the patient thinks it is necessary.
- (7) This examination is not mandatory.

# **3 STUDY OUTCOME VARIABLES**

## 3.1 Performance criteria

## 3.1.1 Primary performance endpoint

The primary performance endpoint is change from baseline in total staining grade according to the Oxford 0-15 grading scheme (corneal staining by fluorescein, nasal and temporal conjunctival staining by lissamine green) at Day 35 in the worst eye.

# 3.1.2 <u>Secondary performance endpoints</u>

Secondary performance endpoints are:

- Change from baseline in total ocular staining grade according to Oxford grading scheme at Day 8 and Day 84 in the worst eye and at Day 8, Day 35 and Day 84 in the contralateral eye;
- Change from baseline in Van Bijsterveld score\* (lissamine green staining) at Day 8, Day 35 and Day 84;
- Change from baseline in DEQ-5 at Day 35 and Day 84;
- Change from baseline in OSDI (Ocular Surface Disease Index) score at Day 8, Day 35 and Day 84;
- Change from baseline in Schirmer test result\* (without anaesthesia) at Day 8, Day 35 and Day 84;
- Change from baseline in TBUT\* (Tear Break-Up Time) at Day 8, Day 35 and Day 84;
- Conjunctival hyperaemia\* using McMonnies photographic scale at Day 8, Day 35 and Day 84;
- HLA-DR (AUF) at Day 84 in Right Eye if eligible eye;
- Objective Scatter Index (OSI) at Day 35 and Day 84;
- Dry Eye symptoms: burning/irritation, stinging/eye pain, itching, eye dryness feeling, foreign body sensation, light sensitivity and fluctuating blurred vision evaluated with a 4-level verbal scale (0 = Absent; 1 = Mild, Present but not disturbing; 2 = Moderate, Disturbing, but not limiting daily activities; 3 = Severe, Very distressing and interfering with daily activities) and change from baseline in total score of Dry Eye symptoms at Day 8, Day 35 and Day 84;
- Performance assessment by the investigator (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory) at Day 35 and Day 84.

#### 3.2 Safety assessments

Other evaluation parameters are:

• Ocular unusual sensation upon instillation at Day 8, Day 35 and Day 84:


<sup>\*</sup>Assessment recorded for each eye will be analysed for the worst eye and the contralateral eye.

Burning/irritation, stinging/eye pain, itching, eye dryness feeling, foreign body sensation, light sensitivity and other symptoms will be graded by the subject according to the following severity scale and with their duration: (0 = Absent; 1 = Mild, Present but not disturbing; 2 = Moderate, Disturbing, but not limiting daily activities; 3 = Severe, Very distressing and interfering with daily activities);

- Far best-corrected visual acuity (in logMAR) at Day 84;
- Tolerance assessment by the patient and the investigator (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory) at Day 35 and Day 84;
- Ocular and systemic adverse events (AE/SAE).

#### 3.3 Derived variables

| Source data | Derivation rule | Label | Format |
|---|---|---|---|
| Possible impact | If screening visit date (SVSTDT for | Possible | 1="Yes" |
| of COVID-19 | VISITNUM=1 in SV table) <= 18MAR2020 | impact of | 0="No" |
| pandemic | Then IMPCOVID=0 | COVID-19 | |
| | | pandemic | |
| | If screening visit date > 18MAR2020 Then | | |
| | IMPCOVID=1 | | |
| Treated eye(s) | If ECLOCLAT = Right eye, Left eye or Both | Safety Set | 1="Yes" |
| at D35 and D84 | eyes at least for one visit among Visit D35 | | 0="No" |
| | and Visit D84, then SS=1 | | |
| | Else SS=0 | | |
| Safety | If SS=1 and DSRANDYN="Y" and at least one | FAS | 1="Yes" |
| population, | post basal value then FAS=1 | population | 0="No" |
| randomized | | | |
| status and post | Else FAS=0 | | |
| baseline | | | |
| performance | Post basal value include: Oxford scores, Van | | |
| evaluations | Bijsterveld scores, DEQ-5 questionnaire, | | |
| | OSDI questionnaire, Schirmer test results, | | |
| | TBUT scores, BCVA, OSI and conjunctival | | |
| | hyperaemia at visit D8, D35 and D84 | | |
| FAS population | If FAS=1 and MAJDEV=0 Then PP=1 | PP | 1="Yes" |
| and major | | Population | 0="No" |
| deviation | Else PP=0 | | |
| | MAJDEV refer to major deviation. All major | | |
| | deviations will be determined during the BR meeting | | |
| Informed | If ICYN = "Y" And SVSTDT Ne "" (Where | Enrolled | 1="Yes" |
| consent signed | Visitnum=1) Then ENROLLED=1 | Population | 0="No" |
| and screen visit | VISIGNAMI-1/ THEN LIVINOLLED-1 | 1 opulation | 0- NO |
| performed | If ICYN Ne "" Or S VSTDT = "" (Where | | |
| periorinea | Visitnum=1) Then ENROLLED=0 | | |
| Oxford 0-15 | To do for both eyes: | Eligible eye | 1="Yes" |
| score, Schirmer | If 4≤0XFGRTOT≤9 And (3≤ SCHIRM≤9 Or .< | Eligible Cyc | 0="No" |
| 30010, 3011111101 | TBUTSUM≤30) Then ELIGEYE=1 | | |
| | 150150WE50) THEN ELIGETE-I | | |

| test and TBUT | Else ELIGEYE=0 | | |
|---|---|---|---|
| total score at D1 | LISC LLIGETE O | | |
| Eligible eyes, | If only one eye is eligible, the eligible eye | Worst eye | 1="Right" |
| Oxford scores, | will be worst eye | Worsteye | 2="Left" |
| Schirmer scores, | will be worst eye | | 2- LCT |
| TBUT total | If both eyes are eligible, then: | | |
| | , - | | |
| scores at D1 | - Eligible eye will be the eye with the | | |
| | worst Oxford score (maximum | | |
| | score of the eyes) | | |
| | - Else If same Oxford score in both | | |
| | eyes, eligible eye will be the eye | | |
| | with the worst Schirmer score | | |
| | (minimum score of the eyes) | | |
| | - Else If same Schirmer score in both | | |
| | eyes, eligible eye will be the eye | | |
| | with the worst TBUT score | | |
| | (minimum score of the eyes) | | |
| | - Else If same TBUT score in both | | |
| | eyes, eligible eye will be right eye. | | |
| | Else If same schirmer score in both eye, | | |
| | eligible eye will be the Right eye | | |
| Worst eye | If WORST=1 Then CONTR=2 | Contralateral | 1="Right" |
| | If WORST=2 Then CONTR=1 | eye | 2="Left" |
| Visit dates at | If DSSTAT="Completed" at the end of the | End of study | DDMMMYYYY |
| Day 84 and | study (visitnum=77, in DS table) Then | date | |
| dates of | ENDDT=SVSTDT where visitnum=5 | | |
| withdrawal | | | |
| | If DSSTAT="Withdrawal" at the end of the | | |
| | study (visitnum=77, in DS table) Then | | |
| | ENDDT=DSENDDT | | |
| Visit dates | FPFV=Min (SVSTDT) where Visitnum=1 | FPFV (First | DDMMMYYYY |
| | | Patient First | |
| | | Visit) | |
| | FPLV= MIN (ENDDT) | FPLV (First | |
| | | Patient Last | |
| | | Visit) | |
| | LPFV=Max (SVSTDT) where Visitnum=1 | LPFV (Last | |
| | | Patient First | |
| | | Visit) | |
| | | , | |
| | LPLV=Max (ENDDT) | LPLV (Last | |
| | | Patient Last | |
| | | Visit) | |
| | | <b>,</b> | |
| | FPR=Min (SVSTDT) where Visitnum=2 | FPR (First | |
| | , | Patient | |
| | | Randomised) | |
| | FPR=Max (SVSTDT) where Visitnum=2 | | |

| | | LDD /L | |
|---|---|---|---|
| | | LPR (Last | |
| | | Patient | |
| | | Randomised) | |
| Visit dates | DURINC=(LPFV-FPFV+1) | Recruitment | Numeric (8.1) |
| | | duration (in | |
| | | days) | |
| LPLV / FPFV | DURSTYM=(LPLV-FPFV +1) /30.44 | Study | Numeric (8.1) |
| , | | duration (in | , , |
| | | months) | |
| Day 1 and Day | BS=Date of D1 | Time | Numeric (8.1) |
| 8, 35 and 84 | SVDELi=(SVSTDATi – BS) | between D1 | ivamene (0.1) |
| visit dates | 378221 (373187111 83) | and Di (in | |
| visit dates | i=Days 9 25 and 94 (data are in line in the | • | |
| | i=Days 8, 35 and 84 (data are in line in the | days) | |
| David viale data | table) | Time to Day | N |
| Day 1 visit date | DTDRYEYE=INPUT(SUBSTR(MHSTDAT, 1, 4), | Time to Dry | Numeric (8.1) |
| and onset date | 8.) | Eye diagnosis | |
| of dry eye | | (in years) | |
| | DEL_DRYEYE=YEAR(BS) – DTDRYEYE | _ | |
| Date of | SVSTDT2=dhms(SVSTDT, 0, 0, SVSTTIM) | Date of Day 1 | DDMMMYYYY |
| randomisation | SVSTDAT (when visitnum=2) | | |
| visit, date and | | Date and | |
| hour of last | When ECCAT="Run-in treatment | time of last | DDMMMYYYY |
| instillation of | compliance": ECENDT2=dhms(ECENDT, 0, 0, | instillation if | HH:MM |
| Hydrabak | ECENTIM) | Hydrabak | |
| Date and time | TIME_HYD_RD= Intck("Hour", ECENDT2, | Time | Numeric (8.1) |
| of | SVSTDT2) | between last | |
| randomisation | | instillation of | |
| and Date and | | Hydrabak | |
| time of last | | and | |
| instillation if | | randomisatio | |
| Hydrabak | | n visit (hours) | |
| Start date of | When ECCAT="Run-in treatment | Treatment | Numeric (8.1) |
| Run-In period | compliance" & ECCSPID in ('1' "): | duration in | (0.2) |
| and End date of | RUNIN DUR= (ECENDT – ECSTDT)+1 | run-in period | |
| Run-In period | | (Hydrabak) | |
| Run in period | | (days) | |
| Treatment | When ECCAT="Run-in treatment | Compliance | 0="No" |
| | | for run-in | 1="Yes" |
| dosage | compliance" & ECCSPID in ('1' "): | | 1- 165 |
| respected | | treatment | |
| during the run- | If ECCOMPYN="N" Then RICOMPL=0 | | |
| in period | If ECCOMPYN="Y" Then RICOMPL=1 | | |
| Start Date of | DURTT=(ECENDT-ECSTDT)+1 | Treatment | Numeric (8.1) |
| Treatment, End | | period (in | |
| Date of | This derivation rule is valid for D1-D35 and | days) | |
| Treatment | D35-D84 periods | | |
| Treatment | DURTT_TOT=SUM(DURTTi) | Total | Numeric (8.1) |
| period (in days) | | treatment | |
| for D1-D35 and | i=D1-D35 and D35-D84 periods | duration (in | |
| D35-D84 | There is one line for D1-D35 period and one | days) | |
| | line for D35-D84 period. Two lines will be | | |

| | summed with SQL procedure in order to | | |
|---|---|---|---|
| | obtain total treatment period (in days) | | |
| Age at Day 1 | If . <age<65 65≤age<85="" agec="3&lt;/td" age≥85="" if="" then=""><td>Age (in classes)</td><td>1="&lt; 65 years"<br/>2="[65; 85<br/>years["<br/>3="≥ 85 years"</td></age<65> | Age (in classes) | 1="< 65 years"<br>2="[65; 85<br>years["<br>3="≥ 85 years" |
| Date of | STUDY DUR D= ENDDT – SVSTDAT (when | Study | Numeric (8.1) |
| Selection visit, Date of withdrawal, | visitnum=1)+1 | duration (in days) | , |
| Mean Daily Dose Regimen at D1-D35 and D35-D84 periods | If ECREGIM="2" INSTILLATIONS/DAY" Then ECREGIMn=2 If ECREGIM="3"INSTILLATIONS/DAY" Then ECREGIMn=3 If ECREGIM="4"INSTILLATIONS/DAY" Then ECREGIMn=4 If ECREGIM ="5" INSTILLATIONS/DAY" Then ECREGIMn=5 If ECREGIM="MORE THAN 5" Then Do If exact number of dose are specified in ECREGIMS Then ECREGIMS Then ECREGIMn=Input(ECREGIMS, 8.) If range of number of dose are specified, Then ECREGIMn=Round(mean of the range, 1) As ECREGIMS is a characters variable, mean | Mean Daily<br>Dose<br>Regimen (n) | Numeric (8.1) |
| | will be calculated individually This derivation rule is valid for D1-D35 and D35-D84 periods | | |
| Oxford total | BSOXFGRTOT=Oxford total score at D1 | Change from | Numeric (8.1) |
| score at Day 1,<br>Oxford Total<br>score of the<br>corresponding<br>eye at Days 8,<br>35 and 84 | (OXFGRTOT) EVOL_OXFGRTOTi=(OXFGRTOTi – BSOXFGRTOT) i=Days 8, 35 and 84 (data are in line in the table) | baseline in<br>Oxford<br>Grading Total<br>score on Day<br>i | |
| and EVOL_ VBGL | · | | · |
| Items of DEQ-5<br>questionnaire at<br>Selection visit,<br>Day 35 and Day<br>84 | If MULTQ51A="" Then DEQ501An=Input(DEQ501A, 8.) If DEQ501A="MISSING%" Or MULTQ51A Ne "" Then DEQ501An=. | DEQ-5-Eye<br>discomfort:<br>How often?<br>(n) | Numeric (8.1) |
| | If MULTQ51B="" Then DEQ501Bn=Input(DEQ501B, 8.) | DEQ-5-Eye<br>discomfort: | |

| <u></u> | | | T |
|---|---|---|---|
| | If DEQ501B="MISSING%" Or MULTQ51B Ne | How intense? | |
| | "" Then DEQ501Bn=. | (n) | |
| | If MULTQ52A="" Then | DEQ-5-Eye | |
| | DEQ502An=Input(DEQ502A, 8.) | dryness: How | |
| | If DEQ502A="MISSING%" Or MULTQ52A Ne | often? (n) | |
| | "" Then DEQ502An=. | , , | |
| | | DEQ-5-Eye | |
| | If MULTQ52B="" Then | dryness: How | |
| | DEQ502Bn=Input(DEQ502B, 8.) | intense? (n) | |
| | If DEQ502B"MISSING%" Or MULTQ52B Ne | interise: (ii) | |
| | "" Then DEQ502Bn=. | סרס ר | |
| | Then DEQ502Bh=. | DEQ-5- | |
| | 15 A 4 11 T O F O 7 " T I | Watery eyes: | |
| | If MULTQ53="" Then | How often? | |
| | DEQ503n=Input(DEQ503, 8.) | (n) | |
| | If DEQ503="MISSING%" Or MULTQ53 Ne "" | | |
| | Then DEQ503n=. | | |
| | This derivation rule is valid for Selection | | |
| | visit, Days 35 and 84 | | |
| | Cases of multi-tick will be discussed during | | |
| | the BR Meeting | | |
| Items of DEQ-5 | If DEQ501An Ne . And DEQ501Bn Ne . And | DEQ-5-Score | Numeric (8.1) |
| questionnaire in | DEQ502An Ne . And DEQ502Bn Ne . And | (n) | |
| numeric format | DEQ503n Ne 1 Then | | |
| at Selection | DEQ5TOT=DEQ501An+DEQ501Bn+DEQ502 | | |
| visit, Day 35 and | An+ DEQ502Bn+DEQ503n | | |
| Day 84 | 7 2.2022 2.2000 | | |
| | This derivation rule is valid for Selection | | |
| | visit, Days 35 and 84 | | |
| | visit, buys 33 und 04 | | |
| | In case of multi-ticked, worst response will | | |
| | be take into account | | |
| DEO E total | | Change from | Numaria (9.1) |
| DEQ-5 total | BSDEQ5TOT= DEQ5TOT at Selection visit | Change from | Numeric (8.1) |
| score at | EVOL_DEQ5TOTi = DEQ5TOTi- BSDEQ5TOT | baseline in | |
| Selection visit, | | DEQ-5 total | |
| DEQ-5 total | i=Days 35 and 84 (data are in line in the | score on Day | |
| score at Day 35 | table) | i | |
| and Day 84 | | | |
| Items of OSDI | If MULTOS1= "" Then | OSDI-Eyes | Numeric (8.1) |
| questionnaire at | OSDI0101n=Input(OSDI0101, 8.) | Sensitive to | |
| Days 1, 8, 35 | If OSDI0101="MISSING%" Or MULTOS1 Ne | Light | |
| and 84 | "" Or OSDI0101="NA" Then OSDI0101n=. | | |
| | | OSDI-Eyes | |
| | If MULTOS2="" Then | Gritty | |
| | OSDI0102n=Input(OSDI0102, 8.) | | |
| | If OSDI0102="MISSING%" Or MULTOS2 Ne | | |
| | ""Or OSDI0102="NA" Then OSDI0102n=. | | |
| I | | | l . |

| | T | | 1 |
|---|---|---|---|
| | If MULTOS12="" | OSDI-Air | |
| | OSDI0112n=Input(OSDI0112, 8.) | Conditioned | |
| | If OSDI0112="MISSING%" Or MULTOS12 Ne | Areas | |
| | "" Or OSDI0112="NA" Then OSDI0112n=. | | |
| | This desiration and is walled for Deve 1 0 25 | | |
| | This derivation rule is valid for Days 1, 8, 35 | | |
| | and 84 | | |
| | Cases of multi-tick will be discussed during | | |
| | the BR Meeting | | |
| | In case of multi-ticked, worst response will | | |
| | , | | |
| | be take into account | | |
| Items of OSDI | OSDI0113b=SUM(OSDI0101n, n, | OSDI- | Numeric (8.1) |
| questionnaire in | OSDI0103n, OSDI0104n, OSDI0105n) | Subtotal | |
| numeric format | | Score | |
| at Days 1, 8, 35 | | Answers 1 to | |
| and 84 | | 5 | |
| 3110 07 | OSDI0114h-SUM/OSDI01065 OSDI01075 | | |
| | OSDI0114b=SUM(OSDI0106n, OSDI0107n, | OCD! | |
| | OSDI0108n, OSDI0109n) | OSDI- | |
| | | Subtotal | |
| | | Score | |
| | | Answers 6 to | |
| | OSDI0115b=SUM(OSDI0110n, OSDI0111n, | 9 | |
| | - | 9 | |
| | OSDI0112n) | | |
| | | OSDI- | |
| | | Subtotal | |
| | This derivation rule is valid for Days1, 8, 35 | Score | |
| | and 84 | Answers 10 | |
| | una 04 | to 12 | |
| Culatatal Casus | NDOCDI Tetal assarbas of assartions | | Numer and a (O. 4) |
| Subtotal Score | NBOSDI=Total number of questions | Number of | Numeric (8.1) |
| Answers 1 to 5, | answered (without NA answered) | questions | |
| OSDI-Subtotal | | answered | |
| Score Answers 6 | | | |
| to 9, OSDI- | OSDITOT=SUM(OSDI0113b,OSDI0114b, | OSDI-Total | |
| Subtotal Score | OSDI0115b) | Sum | |
| | (30101130) | Sum | |
| Answers 10 to | | | |
| 12 at Days 1, 8, | OSDI0118b=(OSDITOT*25)/NBOSDI | OSDI-Total | |
| 35 and 84 | | Score Re- | |
| | | Calculated | |
| | This derivation rule is valid for Days 1, 8, 35 | | |
| | and 84 | | |
| OCDI total sacra | | Change from | Numoric (9.1) |
| OSDI total score | BSOSDI0118b = OSDI0118b at D1 | Change from | Numeric (8.1) |
| at Day 1, OSDI | EVOL_OSDI0118bi = OSDI0118bi- | baseline in | |
| total score at D | BSOSDI0118b | OSDI total | |
| | | score on Day | |
| | i=Days 8, 35 and 84 (data are in line in the | i | |
| | table) | | |
| OSDI total sacra | If 0≤ OSDI0118b <13 then OSDI0118c=1 | OSDI total | 1="Normal" |
| OSDI total score | II 07 O2DIOTTON <12 (HGH O2DIOTT8C=1 | | |
| at Days 1, 8, 35 | | score | 2="Mild" |
| and 84 | If 13≤ OSDI0118b <23 then OSDI0118c=2 | (classes) | 3="Moderate" |
| | | | 4="Severe" |

| | If 23≤ OSDI0118b <33 then OSDI0118c=3 | | |
|---|---|---|---|
| | If 33≤ OSDI0118b ≤100 then OSDI0118c=4 | | |
| | This derivation rule is valid for Days 1, 8, 35 and 84 | | |
| | In statistical results, range of each modality will be specified with footnote | | |
| Schirmer test<br>result at Day 1,<br>Schirmer test<br>result of the<br>corresponding<br>eye at Days 8, | BSSCHIRM= Schirmer test result at D1 (SCHIRM) EVOL_SCHIRMi=(SCHIRMi – BS SCHIRM) i=Days 8, 35 and 84 (data are in line in the table) | Change from<br>baseline in<br>Schirmer test<br>result on Day<br>i | Numeric (8.1) |
| 35 and 84<br>TBUT | MEANTBUT=(TBUT1+TBUT2+TBUT3)/3 | Mean TBUT | Numeric (8.1) |
| measurements 1, 2 and 3 at Days 1, 8, 35 and 84 | This derivation rule is valid for Days 1, 8, 35 and 84 | | |
| Mean TBUT at<br>Day 1, Mean<br>TBUT of the<br>corresponding<br>eye at Days 8,<br>35 and 84 | BSMEANTBUT= Mean TBUT at D1 (MEANTBUT) EVOL_MEANTBUTi=( MEANTBUTi – BS MEANTBUT) i=Days 8, 35 and 84 (data are in line in the table) | Change from<br>baseline in<br>Mean TBUT<br>on Day i | Numeric (8.1) |
| Severity/Intensit<br>y of Dry Eye<br>Symptoms at<br>each visit | If CESEV="ABSENT" Then CESEVn=0 If CESEV="MILD, PRESENT BUT NOT DISTURBING" Then CESEVn=1 If CESEV="MODERATE, DISTURBING, BUT NOT LIMITING DAILY ACTIVITIES" Then CESEVn=2 If CESEV="SEVERE, VERY DISTRESSING AND INTERFERING WITH DAILY ACTIVITIES" Then CESEVn=3 | Severity /<br>Intensity (n) | 0="Absent"<br>1="Mild"<br>2="Moderate"<br>3="Severe" |
| Dry Eye<br>Symptoms | If, for the visit i patient does not have all symptoms, missing symptoms will be created with CESEVn=0 Only for CECAT="Ocular Symptoms" | Severity /<br>Intensity (n) | 0="Absent"<br>1="Mild"<br>2="Moderate"<br>3="Severe" |
| Dry eye<br>symptoms at<br>each visit | SCORE_DES=Sum(CESEVn) Where CECAT=Ocular Symptoms Only for the 7 predefined dry eye symptoms and if the 7 predefined dry eye symptoms are not missing | Total score of<br>Dry Eye<br>symptoms | Numeric (8.1) |

| • | dry eye symptoms are: Burning/Irritation, Sting ody sensation, Light sensitivity and Fluctuating | | ching, Eye dryness |
|---|---|---|---|
| Total score of Dry Eye symptoms at Days 1, 8, 35 and 84 | BS SCORE_DES= Total score of Dry Eye Symptoms at D1 (SCORE_DES) EVOL_SCORE_DESi=(SCORE_DESi- BSSCORE_DES) i=Days 8, 35 and 84 (data are in line in the table) | Change from<br>baseline in<br>total score of<br>dry eye<br>symptoms on<br>Day i | Numeric (8.1) |
| Change from<br>baseline in total<br>score of dry eye<br>symptoms on<br>Day 8 (i.e. Days<br>35 and 84) | If .Z <evol_score_desi<0 evol_score_desci="2" evol_score_desi="" if="" then="">0 Then EVOL_SCORE_DESi&gt;0 Then EVOL_SCORE_DESCi=3 i=Days 8, 35 and 84 (data are in line in the table)</evol_score_desi<0> | Evolution Dry<br>Eye symptom<br>on Day i | 1="Improvemen<br>t"<br>2="Stable"<br>3="Worsening" |
| Symptoms upon instillation | If, for the visit i patient does not have symptoms upon instillation, 6 lines will be created for the 6 predefined symptoms, with CESEVn=0 Only for CECAT="Ocular Symptoms Upon Instillation" | Severity /<br>Intensity (n) | 0="Absent"<br>1="Mild"<br>2="Moderate"<br>3="Severe" |
| Symptoms upon instillation | SCORE_UPON= Sum(CESEVn) Where CECAT= Ocular Symptoms Upon Instillation Only for the 6 predefined dry eye symptoms and if the 6 predefined dry eye symptoms are not missing | Total score of unusual sensation UPON INSTILLATION | Numeric (8.1) |
| • | dry eye symptoms are: Burning/Irritation, Sting ody sensation and Fluctuating blurred vision | ging/Eye pain, Ito | ching, Eye dryness |
| Start of previous and concomitant treatments | If substr(CMSTDAT, 9, 2)="ND" then the day will be replaced by 01 (first day of the month) If substr(CMSTDAT, 6, 5)="ND/ND" then the month and the day will be replaced by 01/01 (first day of the year | Start date of medications (imputed, n) Will be used only to determined type of | DDMMMYYY |
| | Name of the created variable: CMSTDATimp | treatment<br>(previous,<br>concomitant<br>or post-<br>study) | |
| End date of previous and | If substr(CMENDAT, 9, 2)="ND" then the day will be replaced by 28, 30 or 31, depending of the month (last day of the | End date of medication (imputed, n) | |

| concomitant | month) | | |
|---|---|---|---|
| treatments | | Will be used | |
| ti cutilicités | If substr(CMENDAT, 6, 5)="ND/ND" then | only to | |
| | the month and the day will be replaced by | determined | |
| | "12/31" (last day of the year) | type of | |
| | | treatment | |
| | Name of the created variable: | (previous, | |
| | CMENDATimp | concomitant | |
| | | or post- | |
| | | study) | |
| Start date and | If CMSTDT Ne . And CMENDT Ne . Then | Duration of | Numeric (8.1) |
| End date of | PCM_DUR=((CMENDT-CMSTDT)+1)/30.44 | treatment (in | |
| previous and | If CMONGO="Y" Then PCM_DUR=. | months) | |
| concomitant<br>treatments | | | |
| Start date and | If CMSTDATimp Ne . And CMENDATimp Ne . | Duration of | Numeric (8.1) |
| end date of | Then PCM_DUR=((CMENDATimp - | treatment (in | Numeric (0.1) |
| previous and | CMSTDATimp)+1)/30.44 | months, with | |
| concomitant | If CMONGO="Y" Then PCM_DUR=. | imputed | |
| treatments | _ | dates) | |
| Date of | DAKDATD1=Date of instillation at D1 | Date of | DDMMMYYYY |
| Instillation at | (VISITNUM=2) | treatment | |
| Day 1 | | initiation | |
| Date of last | DAKDATLAST=Max(DAKDT) | Date of last | DDMMMYYYY |
| instillation | | treatment | |
| Imputed start | If CMENDAT_dat Ne . And DAKDATD1 Ne . | dispensation Type of | 1="Previous" |
| date and end | And CMENDAT_dat <dakdatd1 .<="" ne="" td=""><td>medication</td><td>2="Concomitant</td></dakdatd1> | medication | 2="Concomitant |
| date of previous | CMTYP=1 | (previous or | " |
| and | | concomitant) | 3="Post-study" |
| concomitant | If CMSTDAT_dat Ne . And DAKDATLAST Ne . | , | , |
| treatment and | And CMSTDAT_dat>DAKDATLAST Then | | |
| date of | CMTYP=3 | | |
| selection visit | | | |
| | If CMENDAT_dat Ne . And DAKDATD1 Ne . | | |
| | And CMENDAT_dat>=DAKDATD1 Then | | |
| | CMTYP=2 | | |
| | In case of ongoing with start date available: | | |
| | If CMTYP=. And CMONGO="Y" And | | |
| | CMSTDAT_dat Ne . And | | |
| | CMSTDAT_dat <dakdatlast td="" then<=""><td></td><td></td></dakdatlast> | | |
| | CMTYP=2 | | |
| | In case of no start date of medication: | | |
| | If CMSTDAT_dat=. And DAKDATD1 Ne . | | |
| | Then CMTYP=2 | | |
| | If no date of treatment initiation: | | |
| | If DAKDATD1=. Then CMTYP=. | | |

| | Medications without type will be reviewed | | |
|---|---|---|---|
| | during the BR Meeting | | |
| HLA-DR at Day 1 and Day 84 | LBHLAREL2=LBHLAREL | HLA-DR<br>positive cells | Numeric (8.1) |
| , | If LBYN="Y" And LBVAL="N" Then | (%, missing | |
| | LBHLAREL2=. | for invalid | |
| | | result) | |
| Tolerance | IF TOLERI In ('SATISFACTORY' | Tolerance | 1="Very |
| assessment by | 'VERY SATISFACTORY') Then TOLERI2=1 | assessment | satisfactory / |
| the investigator | · | by the | Satisfactory" |
| at Day 35 and | If TOLERI In ('NOT VERY SATISFACTORY' | investigator | 2="Not very |
| Day 84 | 'UNSATISFACTORY') Then TOLERI2=2 | | satisfactory / |
| - , - | , | | Unsatisfactory" |
| | This derivation rule is valid for Days 35 and | | , |
| | 84 | | |
| AE start date, | AEDUR=(AEENDT – AESTDT)+1 only if | AE duration | Numeric (8.1) |
| AE end date | AEOUT=" RECOVERED/RESOLVED" | (in days) | |
| AE start date, | AETIME=(AESTDT – DAKDATD1) | AE onset | Numeric (8.1) |
| Start date of | | from First | |
| treatment | | IMD | |
| | | instillation | |
| | | (days) | |
| Start date of | If AESTDT < DAKDATD1 then TEAE=0 | Treatment | 0="No" |
| treatment / | If AESTDT >= DAKDATD1 then TEAE=1 | Emergent | 1="Yes" |
| Time of onset of | | Adverse | |
| AE | In case of missing or uncompleted onset | Event (TEAE) | |
| | date/time, the status will be defined during | | |
| | the Blind Review (BR) meeting according to | | |
| | the information recorded in other fields | | |
| AE type and | If TEAE=1 And localisation in ("BOTH EYES" | Ocular TEAE | 0="No" |
| localisation | "RIGHT EYE" "LEFT EYE") Then OCTEAE=1 | | 1="Yes" |
| | If (TEAE=1 And AELOCLAT="OTHER") Or | | |
| | TEAE=0 Then OCTEAE=0 | | |
| AE type and | If TEAE=1 And AEREL="RELATED" Then | ADE | 0="No" |
| causality | ADE=1 | | 1="Yes" |
| | If TEAE=0 Or (TEAE=1 And AEREL="NOT | | |
| | RELATED") Then ADE=0 | | |
| AE type and | If ADE=1 And AESER ="Y" Then SADE=1 | SADE | 0="No" |
| serious event | | | 1="Yes" |
| | If ADE=0 Or (ADE=1 And AESER="N") Then | | |
| | SADE=0 | | |
| AE type and | If TEAE=1 And AEACN "drug withdrawn" | TEAE leading | 0="No" |
| Action Taken | Then WTEAE=1 | to Medical | 1="Yes" |
| with Study | Else WTEAE=0 | Device | |
| Treatment | | withdrawal | |

# 4 SEQUENCE OF PLANNED ANALYSES

# 4.1 Interim analyses

No interim analysis is planned.

# 4.2 Final analyses and reporting

This SAP described the final statistical analysis.

The analyses will be performed after the database has been cleaned and locked.

A BR meeting will be conducted prior to database lock. Treatment allocations will not be unblinded and no un-blinded analyses will begin until this SAP has been approved by the sponsor.

Any post-hoc exploratory analyses performed to provide support for planned analyses but not identified in this SAP will be documented and reported in appendices to the CSR and clearly identified as unplanned analyses in the text of the CSR.

# 4.3 Changes to statistical information in the clinical trial protocol

In the protocol, the final visit form can either be D84 visit or Withdrawal visit. Withdrawal visits specified in the final visit form will be reviewed during the BR meeting and reclassified to the closest missing planed timepoint (D8, D35 or D84).

Information collected during withdrawal visit will be used in the analysis as reclassified visit.

In the protocol, for the primary performance endpoint, the investigator site and the investigation product-by investigator site interaction was expected to be explored as a secondary analysis prior to presenting the final model. As the number of randomised patients by site is low, investigator site will not be tested but replaced by country effect.

For the primary performance endpoint, additional sensitivity analysis will be performed: Mixed Model for Repeated Measures (MMRM) model will be used including: treatment group, baseline value, visit, treatment group by visit interaction and treatment group by baseline value interaction.

To investigate the bias of recruitment before and after the recruitment interruption, patients will be classified without or with possible impact of COVID-19 pandemic based on their screening visit date respectively up to and including 18 MARS, or after the 18-MAR-2020. Descriptive analysis will be performed according to this variable (populations, countries, premature withdrawal, protocol deviations and demographic characteristics (age and sex). Moreover, for the primary endpoint, an exploratory model will be performed using initial model, adjusted on this new variable.

For the analysis of previous and concomitant medications, ATC level 2 and 4 will be used, instead of level 3 and 4 specified in the protocol.

For performance and tolerance assessment, Wilcoxon signed-rank test will be replaced by Cochran-Mantel-Haenszel (CMH) test, and Chi-2 test for Dry Eye Symptoms will be replaced by Cochran-Mantel-Haenszel (CMH) test.

In the safety endpoints, for the comparison between treatment group of the total score of the 6 predefined symptoms (unusual sensation upon instillation), Student T-test will be performed, instead of the use of Analysis of Covariance (ANCOVA) analysis as specify in the protocol. Student T-test will be performed if the normality of the data is verified. If the data have not normal distribution, Mann-Whitney Wilcoxon test will be used.

#### 5 STATISTICAL METHODOLOGY

# 5.1 Detailed power and sample size

The aim of the study is to demonstrate the non-inferiority of T2259 with regard to Vismed® Multi in terms of performance. The primary performance criterion is the change from baseline of total ocular staining grade in the worst eye on Day 35, evaluated using Oxford 0-15 grading scheme.

As the statistical hypothesis is the non-inferiority of T2259 with regard to Vismed®, the main analysis of the primary criterion will be performed in the Per Protocol population.

A total of 76 patients (i.e. 38 per treatment group) assume at least 90% power to establish the non-inferiority comparison on a one sided two sample t test with  $\alpha$ =2.5 % basis (equivalent to a 95% two sided confidence interval), assuming that the standard deviation is 2.5 and no difference between the 2 groups with a non-inferiority limit set at 2 for the change in total ocular staining grade.

Estimation of the standard deviation and determination of the non-inferiority limit are based upon data of previous studies and literature.

Concerning the non-inferiority limit, according to clinicians, a variation of 2 points in the total Oxford grade, which corresponds to a variation of less than 1 grade in the three areas (corneal, temporal and nasal), is considered as not clinically significant.

For taking into account approximately 15% of patients non—evaluable in Per protocol analysis (premature withdrawals without performance evaluation, patients with major protocol deviation), a total of 90 patients should be randomised in the study.

The non-evaluable patient rate was based on the previous studies major deviations and missing data. For this study, missing data are higher than planned (partially due to Covid-19 pandemia) and the number of randomised patients is 101 to maintain approximately the number of 76 patients evaluable in the Per Protocol.

#### 5.2 Generalities for statistical analyses

After the database lock and the randomisation code release, the statistical analysis will be performed by the statistician of Axonal-Biostatem, using SAS® software v9.4 (GUIDE, SAS Institute, North Caroline, USA), according to this SAP.

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

Disposition and baseline characteristics will be presented overall (globally) and by treatment groups. Performance and safety assessments and exposure/compliance will be presented by treatment groups.

Continuous variables will be summarised using descriptive statistics (number of non-missing data (n), number of missing observations, mean, standard deviation (SD), median, lower quartile (Q1), upper quartile (Q3), minimum and maximum).

Except minimum and maximum, descriptive statistics will be presented with one more decimal than the recorded value.

To compare treatment groups for ordinal qualitative variables, Cochran-Mantel-Haenszel (CMH) test will be used stratified by baseline values (if mentioned), with modified ridit scores and "row mean score differ" option. To compare treatment group when variable will be quantitative, Student T-test will be used, when data distribution will be assumed as normal (Shapiro-Wilk test for normality). If it is not the case, Mann-Whitney Wilcoxon test will be preferred instead.

Quantitative parameters will be also compared between groups using ANCOVA model. Furthermore, the mean change from baseline in total staining grade in the worst eye at Day 35 will be compared between the two treatments based on the MMRM analysis, which assumes:

- Data are Missing At Random (MAR)
- All the available data provide the information about non-observed data
- The treatment effect assume that the withdrawn patients mimic those who continued Assumptions underlying the ANCOVA (respectively MMRM for the sensitivity analysis) will be checked:
  - A histogram of residuals will be plotted to check the assumption of normality
  - The underlying assumptions of normality of residuals will also be checked by using Shapiro-Wilk test
  - Normal probability plot and QQ-plot will be performed to check the assumption of normality
  - Residuals will be plotted against predicted values to check the assumption of heteroscedasticity
  - For ANCOVA models, Levene's test will also be performed to check the homogeneity of variances

For each model (MMRM or ANCOVA) if there is a strong violation of normality assumption, a non-parametric comparison – Wilcoxon Rank Sum Test – will be performed in addition to the initial model.

Frequency distribution (number of non-missing observations (n), count and percentage of each modality,) will be summarized for the categorical variables.

All percentages should be rounded and reported to a single decimal place (xx.x%).

For all variables, the number of missing values will also be reported in the tables, but they will not be counted for the percentage calculation (categorical data).

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

Assessment recorded for both eyes will be presented for the worst eye and for the contralateral eye.

Baseline will be defined as the last value before the first instillation.

Change from baseline is defined as the change from the last assessment before the first instillation of the IMD.

However, if measurements are repeated before and after each instillation, baseline is defined as the assessment before the concerned instillation. In this case, the changes from baseline are defined from values assessed after the IMD intake minus the baseline values (last assessment before concerned IMD).

Time between two dates will be calculated as latest date minus earliest date. Study days prior to first injection date are calculated as (actual date – first injection date), after first injection date as (actual date – first injection date) + 1.

All patient data listings will be edited separately. The subject ID, the concerned eye (Right eye/Left eye), the worst eye (Right eye/Left eye), the treatment group, the visit (if applicable) will be presented as identifier variables. Analysis populations for each patient will appear in all the listings.

All patient data listings described in Section 11.9.2 of Clinical Investigation Report will be edited for all the recorded assessments and derived data by type of parameters: Disposition, Demography, Medical history, Previous and Concomitant treatments, Other baseline characteristics (all assessments recorded only at baseline), Performance assessments and endpoints, Safety examinations – by visit, Adverse event, exposure to treatments (Hydrabak®, T2259, Vismed® Multi), Compliance.

Data listings will be presented sorted by subject ID, eye (if applicable) and timepoint (visit).

All date fields will be presented in a format of ddmmmyyyy (e.g., 01Jan2004) in the listings.

#### 5.3 Multiple Imputations for Handling of Dropouts or Missing data

Treatment Emergent Adverse Events (TEAEs) are AEs that occurred after the first IMD instillation. AEs that occurred the day of the first IMD instillation will be reviewed in detail to identify if AEs appeared before or after the first treatment with IMD (to decide if they have to be considered as TEAEs or not). If no additional information is available, they will be treated as TEAEs.

By default, AEs will be considered as TEAEs if no enough information is available.

For primary analysis performed on FAS, Last Observation Carried Forward (LOCF) method will be applied in case of missing value.

In order to define the type of treatments (previous, concomitant or post-study) and treatment duration, partially start/end dates will be imputed with the following rules for calculations:

#### For treatment start date:

- If only the day is missing, it will be considered as 1<sup>st</sup> for calculations
- If only the year is completed, day and month will be considered as January 1<sup>st</sup> for calculations

#### For treatment end date:

- If only the day is missing, it will be considered as the last day of the month for calculations
- If only the year is completed, day and month will be considered as December 31<sup>st</sup> for calculations

If the date is totally missing, it will not be replaced. Other missing data will not be replaced.

# 5.4 Adjustments for Covariates

For the primary analysis, ANCOVA model will be constructed including investigation product as factor and Oxford total score at baseline (Day1) as continuous covariate.

Country and the investigation product-by country interaction will be in addition explored as a secondary analysis prior to presenting the final model.

Moreover, for the primary endpoint, in MMRM analysis (sensitivity analysis), investigation product, Oxford total score at baseline (Day1), visit, investigation product by visit interaction and Oxford total score at baseline by visit interaction will be in the model.

As sensitivity analysis, for the primary endpoint, possible impact of COVID-19 and investigation product by possible impact of COVID-19 will be added in the ANCOVA model.

There is a single primary performance endpoint in the study (change from baseline in the ocular staining grade at D35 in the worst eye) and non-inferiority will be concluded if it is achieved. Other performance endpoints are defined to be of secondary importance. Thus comparison will be performed at a two-sided significant level of 5% and no adjustment of the type I error will be made.

## 5.5 Multicentre

The investigation was carried out in France, in Spain, in Slovakia and in Poland.

## **6 STATISTICAL ANALYSES**

## 6.1 Study Populations

#### 6.1.1 Protocol Deviations

Protocol deviations will be reviewed during the BR meeting and defined as minor and major deviations. The patients with major deviations will be excluded from the Per protocol population.

The decisions taken by the BR committee will be recorded in the BR meeting minutes.

Furthermore, all minor and major deviations will be recorded in the database: a datafile with all patients and information pertaining to analysis sets and protocol deviations will be created according to BR decisions.

The database will be locked after validation of the BR meeting minutes. A certificate of data lock will be provided, then the blind will be broken, and the analyses will be carried out according to the SAP.

## 6.1.2 <u>Analysis Populations</u>

**Full Analysis Set (FAS)** will be composed of all randomised patients (according to ITT principle, i.e. analysed based on the initial treatment assignment), having used at least one dose of investigation medication and for whom at least one post-baseline performance evaluation will be available.

**Per protocol set (PP)** will be a subset of the FAS without major protocol deviation. The precise reasons for excluding patients from the PP set will be defined and documented before breaking the blind during the BR meeting.

**Safety population (SAF)** will be composed of all patients exposed to the investigation Medical Device, i.e. having used at least one administration of the investigational Medical Device.

Note: Enrolled patients will be patients who have signed the informed consent and for whom the screening visit has been recorded in the e-CRF.

The **Eligible Eye** will be defined by following conditions:

- Oxford 0-15 score  $\geq$  4 and  $\leq$  9 AND;
- At least one of the following objective signs:
  - Schirmer test  $\geq$  3 mm/5 min and  $\leq$  9 mm/5 min, **Or**
  - Sum of 3 TBUT measurements ≤ 30 seconds.
  - o **And** without ophthalmological exclusion criterion

For patient with one eligible eye, this eye is considered as the "Worst eye" (study eye for primary analysis).

For patients with both eligible eyes or no eligible eye, the **Worst Eye** will be:

- Eye with the worst Oxford score;
- If same Oxford score in both eyes: eye with the worst Schirmer score;
- If same Oxford and Schirmer scores in both eyes: eye with the worst TBUT score;
- If same Oxford, Schirmer and TBUT scores in both eyes: right eye.

Note: worse Oxford score means highest value, whereas worse Schirmer score or worse TBUT score means lowest value.

The opposite to the worst eye is the **Contralateral Eye**.

Eligible eyes and Worst eye will be validated during the BR.

## 6.2 Disposition of Patients

Descriptive statistics will be provided. No statistical test will be performed.

- Study dates: first date and last date will be provided for selection visit, inclusion visit and last visit (visit 5 or early withdrawal).
- Number and percentage of patients in each country and each site will be provided in FAS and Safety set.

# Status of patients:

- Among all patients: number and percentage of patients selected and not selected, reason if not selected (as reported by the investigator at the selection visit)
- Among selected patients: number and percentage of patients who attended inclusion visit, number and percentage of patients included and not included, reason if not included (as reported by the investigator on end-of-study page: Adverse event, lack of performance, withdrawal by subject, lost to follow-up, screen failure, other)
- Among included patients: randomised (Yes, No)
- Among randomised patients: number and percentage of patients with visits done (for each visit: Yes, No), visit type if Visit 5 done (Day 84 +/-7 days, Premature discontinuation visit), has the patient completed the study (Yes, No), reason if study not completed (Adverse event, lack of performance, withdrawal by subject, lost to follow-up, screen failure, other)

Non-selected patients, non-included patients and early withdrawals will be individually listed.

Note: In case of withdrawal, withdrawal visit will be re-assigned depending to the date of withdrawal. The withdrawal visit will be re-assigned to the closest planned missing visit (D8, D35 or D84). All re-assigned withdrawal visits will be discussed during BR and recorded in the BR meeting minutes.

#### Analysis sets:

- From randomised patients: Number and percentage in safety population, number and percentage of patients excluded from safety population and reason(s) for exclusion
- From safety population: Number and percentage in FAS, number and percentage of patients excluded from FAS and reason(s) for exclusion
- From FAS: Number and percentage in PP, number and percentage of patients excluded from PP and reason(s) for exclusion
- Number and percentage of patients with major and minor protocol deviations, globally and for each section of deviation (inclusion criteria deviation, exclusion criteria deviation, randomisation, visit windows and chronology, run-in treatment compliance, IMD compliance, primary performance endpoint and secondary efficacy endpoints, other), in FAS.


Minor and major deviations will be individually listed, an exhaustive data listing of all patients and information pertaining to analysis sets will also be provided.

Time between visits: time from inclusion visit will be described at selection visit and post-inclusion visits in FAS. For time between randomisation (inclusion) visit date and selection visit date: Randomisation visit date (Day 1) – Selection visit date. For Day 8, Day 35 and D84 it will be calculated as follow: D8 / D35 / D84 visit date – Randomisation visit Date (Day 1).

Time from inclusion visit to Visit 5 will be provided separately for patients for whom visit 5 = Day 84 +/7 days and for patients for whom Visit 5 is a premature discontinuation visit.

Study duration will be described in FAS.

Patients accountability will be described thanks to the flowchart below:



## 6.3 Demographic and Baseline Characteristics

Parameters below will be described globally and by treatment group on PP population and FAS, and Safety population if it differs from FAS.

- Demographic data
  - Sex
  - Age
  - Age in classes (<65 years old, >=65 and < 85 years old, >= 85 years old)
- Baseline characteristics (at selection and randomization visits) will be displayed in the performance tables, as described in the Section 6.7.
- History of dry eye
  - o Time from the Dry eye diagnosis (calculated at selection visit)
  - Aetiology of the dry eye (primary/secondary Sjögren syndrome/Meibomian gland deficiency/Non-Sjögren aqueous deficiency/other)
     A listing of other aetiology will be produced.
  - Eligible eye (none/right eye/left eye/both eyes)
  - Worse eye (right eye/left eye)

# - Medical and surgical history

Medical and surgical history has been coded with MedDRA dictionary (version 22.0).

The number and percentage of patients experiencing at least one medical or surgical history will be provided, overall and by MedDRA primary SOC and PT, separately for ocular medical history other than the studied disease, ocular surgery history other than the studied disease and systemic surgery history other than the studied disease.

Note: Results will be provided by descending frequency (for SOCs and for PTs within SOC, for the whole population analysed)

## 6.4 Subgroup analysis

Patients will be classified without or with possible impact of COVID-19 pandemic based on their Selection visit date respectively up to and including 18-MARS-2020, or after the 18-MAR-2020. The following summaries will be performed:

- Number (%) of patients in each analysis set and reasons for exclusion by possible impact of COVID19
- Number (%) of patients in each country by possible impact of COVID-19
- Number (%) of premature withdrawal by possible impact of COVID-19
- Protocol deviations by possible impact of COVID-19
- o Demographic characteristics by possible impact of COVID-19

Analysis sets will be presented on all randomised subjects, protocol deviation on FAS population, whereas countries, premature withdrawal and demographic characteristics will be presented on FAS and SAF populations.

# 6.5 Previous, Concomitant and Post-Study Medications

Previous and concomitant medication will be described overall and by treatment group in the FAS and the PP, separately for ocular and non-ocular treatments.

Treatments have been coded using the WHO Drug Dictionary Enhanced (WHODrug: B3 Global 2018Q3)

Number and percentage of patients with at least one previous or concomitant treatment will be presented overall and by ATC classification level 2 and ATC classification level 4, according to the 3 observation periods:

- Previous treatments: Treatments ended before the first instillation of the IMD or the same day
- Post-study treatment: Treatments started after the last instillation of IMD or the same day
- Concomitant treatments: Treatments started between the first and last instillation of the IMD (or the same day) or treatments started before the first instillation of the IMD and ended after the first instillation of the IMD.

Note: Results will be provided by descending frequency (for ATC classification level 2 and ATC classification level 4 with level 2, for the whole population analysed)

The Individual data listing will present all CRF items and calculated variables as treatment duration and periods (previous, post-study or concomitant treatment).

# 6.6 Treatment exposure and compliance

The following variables will be described by treatment group, in the Safety population, the FAS and the PP, without performing any statistical test:

- Treatment duration in run-in period (Hydrabak) (days): quantitatively
  - = Date of the last instillation of Hydrabak Date of the first instillation of Hydrabak + 1
- Time between last instillation of Hydrabak and inclusion visit date (hours): quantitatively
- Run-in treatment compliance: dosage for Hydrabak respected? (Yes, No)
- Study treatment duration (days): quantitatively, for the whole study and separately for D1-D35 and D35-D84 periods
- Mean daily dose regimen: quantitatively and in classes (0, 1, 2, 3, 4, 5, >5) during all the study and separately for D1-D35 and D35-D84 periods

When dose regimens are equal to "more than 5 instillation/days", it will be reviewed and converted into numeric values. In case of range, mean range value rounded to the integer will be used. Patients without any treated eye will have 0 for the mean daily dose regimen.
Patients for whom mean daily dose regimen was different from 2 to 4 instillations/day will be individually listed (treatment dates at each visit, mean daily regimen, comments).

## 6.7 Performance analyses

## 6.7.1 Primary Performance Endpoint

Primary performance endpoint will be analysed only in the worst eye.

Descriptive tables will be produced presenting selection, baseline (D1), Day 8, Day 35 and Day 84 Oxford Total score and change from baseline for Oxford Total score at Day 8, Day 35 and Day 84.

Oxford grade at each visit and change from baseline at Day 8, Day 35 and Day 84 will be also described for each panel: temporal bulbar conjunctiva, corneal area and nasal bulbar conjunctiva.

The hypothesis of non-inferiority of T2259 compared to Vismed Multi will be tested by calculating the bilateral 95% CI of the difference between groups (T2259 – Vismed Multi) of the change from baseline of Oxford Total Score on Day 35. A two-way analysis of covariance (ANCOVA) model will be constructed using main effects of investigation product and baseline score as covariate. Adjusted means by investigation product will be presented as well as an estimate of the difference between adjusted means.

A 95% two-sided confidence interval, based on the ANCOVA model (2), will be computed for the difference of T2259 minus Vismed Multi. If the upper bound is no higher than 2 points for the PP population, it will be concluded that the null hypothesis can be rejected and that T2259 is non-inferior to Vismed Multi.

The result will be presented as follow:

| Population | T2259<br>(N=XX) | Vismed®<br>Multi<br>(N=XX) | Difference<br>T2259 – Vismed<br>Multi | SE of<br>Difference<br>T2259 –<br>Vismed<br>Multi | 95% CI |
|---|---|---|---|---|---|
| Day 1 (baseline) mean (SD) | X1 | Y1 | | | |
| Day 35 mean (SD) | X2 | Y2 | | | No. |
| Adjusted mean change<br>(SE) between Day 1 and<br>Day 35 | [X2-<br>X1]*(SE) | [Y2-Y1]*(SE) | [X2-X1] -[Y2-Y1] | SE | [ Min - <b>Max**]</b> |

<sup>\*</sup> These values were expected as negative, meaning an improvement of the Oxford score.

This analysis will be performed firstly on the Per Protocol population on the observed data.

Same analysis will be performed on FAS population with imputation of values in case of missing data with LOCF technique (Day 8 or value in case of withdrawal) and without imputation (observed cases) for confirmation.

<sup>\*\*</sup> The upper bound indicates the maximal difference of change in disfavour of T2259.

The country and the investigation product-by-country interaction will be explored as a secondary analysis prior to presenting the final model (1).

Same analysis as principal analysis (ANCOVA model) will be performed adjusted on possible impact of COVID-19 pandemic (3).

Another sensitivity analysis will be performed using MMRM model (4). This model will be constructed using main effects of investigation product and visit as factors and total Oxford baseline score as continuous covariate. Interactions between treatment and visit, treatment and baseline total Oxford score will also be included. REML method will be used and the covariance structure will be defined as unstructured: unstructured approach makes no assumption about the correlations among visits. If the analysis fails to converge, then spatial covariance, compound symmetry, or first order autoregressive model (A1) structure will be used. The best model fit will be determined by the AIC.

For the ANCOVA and MMRM analyses, the following MIXED procedure (SAS®) will be used.

| Model | Method | SAS code |
|-------|--------|---------------------------------------------------|
| (1) | ANCOVA | PROC MIXED DATA=XX ORDER=DATA; |
| . , | | WHERE PP = $1$ ; /* OR FAS=1 */ |
| | | CLASS TT COUNTRY; |
| | | MODEL EVOL = TT BASELINE COUNTRY TT*COUNTRY / |
| | | SOLUTION ALPHA=0.05; /* OTHER CHARACTERISTICS CAN |
| | | BE ADDED HERE */ |
| | | LSMEANS TT / DIFF=CONTROL CL OM; |
| | | RUN; |
| (2) | ANCOVA | Final model: |
| | | PROC MIXED DATA=XX ORDER=DATA; |
| | | WHERE PP = 1; $/*$ OR FAS=1 */ |
| | | CLASS TT; |
| | | MODEL EVOL = TT BASELINE / SOLUTION ALPHA=0.05; |
| | | /* OTHER CHARACTERISTICS CAN BE ADDED HERE */ |
| | | LSMEANS TT / DIFF=CONTROL CL OM; |
| | | RUN; |
| (3) | ANCOVA | PROC MIXED DATA=XX ORDER=DATA; |
| , , | | WHERE PP = $1$ ; /* OR FAS=1 */ |
| | | CLASS TT COVID; |
| | | MODEL EVOL = TT BASELINE COVID TT*COVID/ SOLUTION |
| | | ALPHA=0.05; /* OTHER CHARACTERISTICS CAN BE ADDED |
| | | HERE */ |
| | | LSMEANS TT / DIFF=CONTROL CL OM; RUN; |
| | | RON, |
| (4) | MMRM | PROC MIXED DATA=XX METHOD=REML; |
| | | WHERE PP=1; /* OR FAS=1 */ |
| | | CLASS TT SUBJID VIS; |
| | | MODEL EVOL = TT VIS BASELINE TT*VIS |
| | | BASELINE*VIS / DDFM=SATTERTH SOLUTION |
| | | ALPHA=0.05; |
| | | REPEATED VISIT / TYPE=UN SUBJECT=SUBJID; |
| | | LSMEANS TT*VIS / PDIFF CL; |

```
ESTIMATE "D35 (VISIT 4) - DIFF T2259 - VISMED"
TREATMENT 1 -1
VISIT*TT 0 1 0 0 -1 0 / CL;
ODS OUTPUT LSMEANS=MEANS DIFFS=DIF;
RUN;
```

### 6.7.2 <u>Secondary Performance Endpoints</u>

Secondary performance endpoints analysis will be provided in the PP population and the FAS population and for both worse eye and contralateral eye.

#### Oxford total score

Descriptive summaries for the Oxford Total score, change from baseline and summaries by panel will be repeated for the contralateral eye in the same manner as for the Primary Endpoint analysis.

Change from baseline in Oxford total score at D8 and D84 on worst eye and at D8, D35 and D84 in contralateral eye will be analysed using an ANCOVA model, constructed using main effects of investigation product and baseline score as covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 – Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

Van Bijsterveld score\* (lissamine green staining)

All items used to calculate the total score will be tabulated, by treatment group, with frequency and percentage at each time point (Selection visit, D1, D8, D35 and D84). Total score and change from baseline will be tabulated, by treatment group, with all parameters specified in part 7.3 (quantitative variables). These analyses will be performed at Day 8, Day 35 and Day 84 on both worst and contralateral eye.

Change from baseline in Van Bijsterveld total score at D8, D35 and D84 for both worst and contralateral eye will be analysed using an ANCOVA model, constructed using main effects of investigation product and baseline score as covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 – Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

\*Assessment recorded for each eye will be analysed for the worst eye and the contralateral eye.

#### DEQ-5 total score

Each question (1a, 1b, 2a, 2b and 3) will be presented, by treatment group, by frequency and percentage at each time point (Selection visit, D35 and D84). Total score and change from baseline will be tabulated, by treatment group. These analyses will be performed at Day 35 and Day 84.

Change from baseline in DEQ-5 total score at D35 and D84 will be analysed using an ANCOVA model, constructed using main effects of investigation product and baseline score as

covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 – Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

- OSDI (Ocular Surface Disease Index) total score

Each question (from Q1 to Q12) will be presented, by treatment group, by frequency and percentage at each time point (D1, D8, D35 and D84). Total score and change from baseline will be tabulated, by treatment group. These analyses will be performed at Day 8, Day 35 and Day 84.

Change from baseline in OSDI total score will be analysed at D8, D35 and D84 using an ANCOVA model, constructed using main effects of investigation product and baseline score as covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 – Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

Moreover, at each time point, OSDI total score will be presented, by treatment group, by frequency and percentage with the following modalities: Normal ([0-13[), Mild ([13-23[), Moderate ([23-33[) and Severe ([33-100]) and Cochran-Mantel-Haenszel (CMH) test will be performed for D35 and D84.

- Schirmer Test result\* (without anaesthesia)

Schirmer test results at each time point (D1, D8, D35 and D84) and change from baseline will be tabulated, by treatment group. These analyses will be performed at Day 1, Day 8, Day 35 and Day 84 on both worst and contralateral eye.

Change from baseline in Schirmer Test result will be analysed at D8, D35 and D84 on both worst and contralateral eye using an ANCOVA model, constructed using main effects of investigation product and baseline score as covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 – Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

\*Assessment recorded for each eye will be analysed for the worst eye and the contralateral eye.

TBUT\* (Tear Break-Up Time)

Each measure of TBUT will be presented, by treatment group, by frequency and percentage at each time point. Mean TBUT at each time point (D1, D8, D35 and D84) and change from baseline will be tabulated, by treatment group for both worst and contralateral eye. These analyses will be performed at Day 8, Day 35 and Day 84.

Change from baseline in mean TBUT will be analysed at D8, D35 and D84 on both worst and contralateral eye using an ANCOVA model, constructed using main effects of investigation product and baseline score as covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 – Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

- Conjunctival hyperaemia\* using McMonnies photographic scale

Score of Conjunctival hyperaemia will be tabulated, by treatment group, at each time point

(D1, D8, D35 and D84) using frequency and percentage. Treatment groups will be compared using a Cochran-Mantel-Haenszel (CMH) test based on modified ridit scores (using SCORES=MODRIDIT option in FREQ procedure), stratified by the baseline value.

\*Assessment recorded for each eye will be analysed for the worst eye and the contralateral eye.

# Dry eye symptoms

Each Dry Eye symptom at Day 8, Day 35 and Day 84 will be compared between treatment group using percentage of patient with an improvement, a stability or a degradation from baseline using a Cochran-Mantel-Haenszel (CMH) test.

Total score and change from baseline will be tabulated, by treatment group. These analyses will be performed at Day 8, Day 35 and Day 84.

Change from baseline in Dry Eye Symptoms total score will be analysed at D8, D35 and D84 using an ANCOVA model, constructed using main effects of investigation product and baseline score as covariate. The LS ("adjusted") means for each treatment arm and estimates of the difference between groups (T2259 — Vismed® Multi) will be presented along with the respective two-sided, 95% CI. Two-sided p-values will be presented for the treatment difference.

#### - Performance assessment

Performance assessment by the investigator will be described by treatment group at Day 35 and Day 84 in 4 classes. An additional description will be provided in 2 classes (Very satisfactory or satisfactory, not very satisfactory or unsatisfactory). Comparison between groups on performance assessment in 4 classes will be performed using a Cochran-Mantel-Haenszel (CMH) test.

For OSI score, only listing will be provided with all corresponding items CRF.

For HLA-DR, quantification (AUF) and percentage will be presented on the whole population. Added analysis will be performed on patients with severe dry eye (OSDI>33 and/or Corneal Fluorescein Staining  $\geq$  3 at the baseline visit).

### 6.8 Safety Analysis

Safety endpoints and adverse events analysis will be provided in the Safety population by treatment group as received.

## 6.8.1 Safety endpoints

- Descriptive tables will be produced by frequency and percentage, for the presence of each ocular unusual sensation UPON INSTILLATION at least one time during the study (for each ocular unusual sensation UPON INSTILLATION)
- Descriptive tables will be produced by frequency and percentage, for each ocular unusual sensation UPON INSTILLATION and by mean (SD) for the total score for the 6 predefined symptoms at Day 8, Day 35 and Day 84.
- The total score for the 6 predefined symptoms will be compared between treatment groups using Student T-test, if data have normal distribution. If it is not the case, Mann-Whitney Wilcoxon test will be used.

Note: For the analysis of ocular unusual sensation UPON INSTILLATION, usual severity, usual duration and frequency will be set to 0 if the patient felt no ocular unusual sensation upon instillation or if the severity is equal to 0 (absent).

- Far best-corrected visual acuity (in logMAR) at Selection visit, Day 35 and Day 84 will be described by mean (SD) for the worst eye and for the contralateral eye. The frequency distribution will be also presented in /10 (1/10, 2/10 to 10/10, >10/10);
- Tolerance assessment by the investigator and by the patient at Day 35 and Day 84 will be described in 4 classes and in 2 classes (Very satisfactory or satisfactory, not very satisfactory or unsatisfactory). The treatment groups for 4 classes description will be compared using a Cochran-Mantel-Haenszel (CMH) test.

# 6.8.2 Adverse events

The adverse events were coded using the MedDRA dictionary version 22.0.

Treatment-emergent AEs (TEAEs) will be defined as AEs with onset date on or after the first day of the IMD instillation. If the AE onset date is not available, AEs will be considered as TEAEs by default.

Ocular and systemic AEs will be analysed separately on the basis of the localisation as recorded by the investigator in the CRF, i.e., localisation = Right eye, Left eye or Both eyes for ocular TEAEs, and localisation = Other for non-ocular TEAEs.

The number and percentage of patients experiencing at least one TEAE will be provided by treatment group, overall by MedDRA primary SOC and PT, for the following categories of adverse events:

- All TEAEs;
- Non-serious TEAEs;
- Treatment related TEAEs (i.e. related or missing relationship with the IMD);
- Serious TEAEs;
- TEAEs leading to medical device withdrawal.
- TEAEs by severity
- TEAEs by relationship with the IMD

Note: Results will be provided by descending frequency (for SOCs and for PTs within SOC, for the whole population analysed).

Individual patient data listings of AEs will be performed for overall AEs, SAEs and SADEs, separately for ocular and systemic AEs. The following variables will be presented:

Treatment group,

- Patient's identifier.
- Worse eye (right eye / left eye)
- Dry eye aetiology
- Gender,
- Age at baseline (Day 1),
- Diagnosis (verbatim),
- SOC,
- PT,
- Localisation,
- Date / time of occurence,
- Time to occurence (days) from the date of the first IMD instillation,
- Treatment-emergence
- Date / time of recovery / date of death, if any,
- Duration (days),
- Outcome,
- Frequency and details,
- Severity,
- Action taken regarding the IMD,
- Requirement for therapy adjustment / modification,
- Requirement for surgical / medical procedure,
- Seriousness,
- Relationship with the IMD in the investigator's opinion,
- Relationship with protocol procedure.

Listings will be sorted by treatment group, patient's identifier and date of onset.

The Individual data listing will present all CRF items and calculated variables as TEAE (Yes/No), time between first instillation of the study and the start date, time between first instillation and stop date, duration of the adverse event.

Listing of Deaths, Other Serious adverse events, discontinuations due to adverse events and other adverse events of special interest will be also provided for narratives.

Discontinuations due to adverse events include drug related AE leading to premature IMP drug OR study withdrawal (i.e. drug related AE with action taken = drug withdrawn OR End of study with premature discontinuation due to this AE) will be listed.

Patient data listings of COVID-19 AEs (PT: COVID-19, Coronavirus infection) will also be produced.

Individual patient data listings of non-emergent AEs will be performed on the SAF population, separately for ocular and systemic AEs.

A excel file with relevant information will also be performed for the CSR narrative.

### 6.8.3 Device deficiencies

Not applicable.

### 7 REPORTING CONVENTIONS

#### 7.1 Software used

Statistical analysis will be made using SAS® GUIDE software (version 9.4). Tables results will be computed with SAS® GUIDE software (version 9.4). Figures will be created using Microsoft® Excel or SAS®GUIDE version 9.4.

#### 7.2 General considerations

All p-values will be rounded to 3 decimal places. If a rounded p-value is 0.000 (i.e., the actual p-value is less than 0.0005), then this will be presented as a p-value of "<0.001". All date fields will be presented in a format of ddmmmyyyy (e.g., 01Jan2004) in the listings.

# 7.3 Statistical summary conventions

For tables, sample sizes for each treatment group will be presented as total in the column header (N=xxx), where appropriate. Sample sizes shown with summary statistics are the number (n) of patients with non-missing values.

Summaries for categorical variables will include only categories that patients had a response in. Percentages corresponding to null categories (cells) will be suppressed. All summaries for continuous variables will include: N, N missing, mean, SD, median, Q1-Q3, minimummaximum and 95%CI. All percentages should be rounded and reported to a single decimal place (xx.x%). If percentages are reported as integers, percentages greater than 0% but <1% will be reported as <1%, whereas percentages greater than 99% but <100% will be reported as >99%. A percentage of 100% will be reported as 100%. No value of 0% should be reported. Any computation of percent that results in 0% is to be reported as a blank.

# 7.4 Examples of tables, listings and figures

# 7.4.1 Quantitative variables

Table xx: Description of quantitative variables

| | | T2259<br>N=xxx | Vismed<br>N=xxx | Total<br>N=xxx | p-value |
|---|---|---|---|---|---|
| Variable 1 | N | Х | X | Х | |
| | Mean ± SD | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | x.xxxx |
| | Median | XX.X | XX.X | XX.X | |
| | 95%CI | [xx.xx; xx.xx] | [xx.xx; xx.xx] | [xx.xx; xx.xx] | |
| | Q1 ; Q3 | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | |
| | Min.; Max. | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | |
| | Missing | Х | X | X | |
| Variable 2 | N | Х | Х | Х | |
| | Mean ± SD | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | x.xxxx |

| | T2259<br>N=xxx | Vismed<br>N=xxx | Total<br>N=xxx | p-value |
|-------------|----------------|-----------------|----------------|---------|
| Median | xx.x | XX.X | XX.X | • |
| 95%CI | [xx.xx; xx.xx] | [xx.xx; xx.xx] | [xx.xx; xx.xx] | |
| Q1 ; Q3 | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | |
| Min. ; Max. | xx.xx; xx.x | xx.xx; xx.x | xx.xx; xx.x | |
| Missing | Х | Х | X | |

Total column will be presented only for patients' disposition and for baseline characteristics.

# 7.4.2 Qualitative variables

Table xx: Description of qualitative variables

| | | T2259<br>N=xxx | | Vismed<br>N=xxx | | p-value |
|---|---|---|---|---|---|---|
| | | N (%) | 95%CI | N (%) | 95%CI | |
| Variable 1 | N | x | | x | | |
| | Missing | х | | X | | |
| | Modality 1 | xx (xx.x%) | [xx.x; xx.x] | xx (xx.x%) | [xx.x; xx.x] | x.xxx |
| | <b>Modality 2</b> | xx (xx.x%) | [xx.x; xx.x] | xx (xx.x%) | [xx.x; xx.x] | |
| Variable 2 | N | х | | Х | | |
| | Missing | х | | X | | |
| | Modality 1 | xx (xx.x%) | [xx.x; xx.x] | xx (xx.x%) | [xx.x; xx.x] | X.XXX |
| | <b>Modality 2</b> | xx (xx.x%) | [xx.x; xx.x] | xx (xx.x%) | [xx.x; xx.x] | |

Table xx: Number (%) of patients selected/not selected and reasons in case of non-selection – All screened patients

| | | Total<br>N=XX |
|-------------------------|----------|------------------------|
| Selected patient | N | Х |
| | No | X <sub>1</sub> (XX.X%) |
| | Yes | X (XX.X%) |
| Reason of non-selection | N | $X_1$ |
| | Reason 1 | X (XX.X%) |
| | Reason 2 | X (XX.X%) |
| | Reason n | X (XX.X%) |

Table xx: Number (%) of patients at each visit and type of last visit – Randomised patients

| | | T2259<br>N=xxx | Vismed<br>N=xxx | Total<br>N=XX |
|---|---|---|---|---|
| Selection visit performed | N | Х | Х | Х |
| | No | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Yes | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| D8 visit performed | N | x | Х | Х |
| | No | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Yes | X (XX.X%) | X (XX.X%) | X (XX.X%) |

|------------------|--------------|--------------|
|------------------|--------------|--------------|

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

| D35 visit performed | N | Χ | Χ | Χ |
|---|---|---|---|---|
| | No | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Yes | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| D84 visit performed | N | X | Χ | Х |
| | No | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Yes | X <sub>1</sub> (XX.X%) | X <sub>1</sub> (XX.X%) | X <sub>1</sub> (XX.X%) |
| Type of D84 visit | N | $X_1$ | $X_1$ | X <sub>1</sub> |
| | D84 visit | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Withdrawal visit | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Table xx: Number (%) of patients in each populations and reasons of exclusion – Randomised patients

| | T2259<br>N=xxx | Vismed<br>N=xxx | Total<br>N=XX |
|---|---|---|---|
| N | Х | Х | Χ |
| No | X <sub>0</sub> (XX.X%) | X <sub>0</sub> (XX.X%) | X <sub>0</sub> (XX.X%) |
| Yes | X <sub>1</sub> (XX.X%) | X <sub>1</sub> (XX.X%) | X <sub>1</sub> (XX.X%) |
| N | $X_0$ | $X_0$ | $X_0$ |
| Reason 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Reason 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Reason n | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| N | $X_1$ | $X_1$ | $X_1$ |
| No | X <sub>2</sub> (XX.X%) | X <sub>2</sub> (XX.X%) | X <sub>2</sub> (XX.X%) |
| Yes | X <sub>3</sub> (XX.X%) | X <sub>3</sub> (XX.X%) | X <sub>3</sub> (XX.X%) |
| N | $X_2$ | $X_2$ | $X_2$ |
| Reason 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Reason 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Reason n | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| N | X <sub>3</sub> | <b>X</b> <sub>3</sub> | X <sub>3</sub> |
| No | X <sub>4</sub> (XX.X%) | X <sub>4</sub> (XX.X%) | X <sub>4</sub> (XX.X%) |
| Yes | X <sub>5</sub> (XX.X%) | X <sub>5</sub> (XX.X%) | X <sub>5</sub> (XX.X%) |
| | No Yes N Reason 1 Reason 2 Reason n N No Yes N Reason 1 Reason 2 Reason n | N X No X <sub>0</sub> (XX.X%) Yes X <sub>1</sub> (XX.X%) N X <sub>0</sub> Reason 1 X (XX.X%) Reason 2 X (XX.X%) Reason n X (XX.X%) N X <sub>1</sub> No X <sub>2</sub> (XX.X%) Yes X <sub>3</sub> (XX.X%) N X <sub>2</sub> Reason 1 X (XX.X%) Reason 2 X (XX.X%) Reason n X (XX.X%) N X <sub>3</sub> No X <sub>4</sub> (XX.X%) | N X X No X <sub>0</sub> (XX.X%) X <sub>0</sub> (XX.X%) Yes X <sub>1</sub> (XX.X%) X <sub>1</sub> (XX.X%) N X <sub>0</sub> X <sub>0</sub> Reason 1 X (XX.X%) X (XX.X%) Reason 2 X (XX.X%) X (XX.X%) N X <sub>1</sub> X <sub>1</sub> No X <sub>2</sub> (XX.X%) X <sub>2</sub> (XX.X%) Yes X <sub>3</sub> (XX.X%) X <sub>3</sub> (XX.X%) N X <sub>2</sub> X <sub>2</sub> Reason 1 X (XX.X%) X (XX.X%) N X <sub>2</sub> X <sub>2</sub> Reason 2 X (XX.X%) X (XX.X%) N X <sub>3</sub> X <sub>3</sub> No X <sub>4</sub> (XX.X%) X <sub>4</sub> (XX.X%) |

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

| Reason of exclusion of PP population | N | $X_4$ | $X_4$ | $X_4$ |
|---|---|---|---|---|
| | Reason 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Reason 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | <br>Reason n | X (XX.X%) | X (XX.X%) | X (XX.X%) |

# 7.4.3 <u>Protocol deviations</u>

Table xx: Protocol deviations – XX population

| | T2259 | Vismed | Total |
|-------------------------------|-------------|-------------|-------------|
| | N=xxx | N=xxx | N=xxx |
| At least one major deviation | | | |
| Deviation 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Deviation 2 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| At least one minor deviation* | | | |
| Deviation 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Deviation 2 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Only minor deviation | | | |
| Deviation 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Deviation 2 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

<sup>\*</sup> includes major deviations

# 7.4.4 Adverse Events

Table xx: Overview of (\*) TEAEs – Safety population

| | T2259 | Vismed |
|-------------------------------|-------------|-------------|
| | N=xxx | N=xxx |
| Any TEAE | xx (xx.x %) | xx (xx.x %) |
| Any serious TEAE | xx (xx.x %) | xx (xx.x %) |
| Any IMP-related TEAE | xx (xx.x %) | xx (xx.x %) |
| Any TEAE leading to premature | xx (xx.x %) | xx (xx.x %) |
| IMD withdrawal | | |

Programming notes: replace (\*) by "ocular" and "systemic"

Table xx: AEs description by SOC and PT

| | | T2259 | | | Visme | ed |
|--------------------------------|-------|-------|------|-----|-------|------|
| SOC and PT | N=xxx | | | | N=xx | x |
| | ΑE | n | % | ΑE | n | % |
| | (1) | (2) | (3) | (1) | (2) | (3) |
| Patients with at least one (*) | XX | xx | XX.X | XX | XX | XX.X |

| SOC and PT | T2259<br>N=xxx | | | | Visme<br>N=xx | |
|---|---|---|---|---|---|---|
| | AE<br>(1) | n<br>(2) | %<br>(3) | AE<br>(1) | n<br>(2) | %<br>(3) |
| SOC 1 | XX | XX | xx.x | XX | XX | XX.X |
| SOC 1 – PT 1 | XX | XX | xx.x | XX | XX | xx.x |
| SOC 1 – PT 2 | XX | XX | XX.X | XX | XX | xx.x |
| | XX | XX | XX.X | XX | XX | xx.x |
| SOC 2 | XX | XX | XX.X | XX | XX | xx.x |
| SOC 2 – PT 1 | XX | XX | XX.X | XX | XX | xx.x |
| SOC 2 – PT 2 | XX | XX | XX.X | XX | XX | xx.x |
| | XX | XX | XX.X | XX | XX | xx.x |

- (1) Number of AEs: each AE is counted only once per SOC/PT
- (2) Number of subjects with at least one AE: each patient is counted only once per SOC/PT
- (3) % of subjects with at least one AE

MedDRA version 22.0

SOC=System Organ Class, PT=Preferred Term, AE=Adverse Event.

Programming notes: replace (\*) by TEAE, ADE or SAD, depending on the table; when needed, update abbreviations.

Table xx: All TEAEs by SOC, PT and severity (XX treatment group) – Safety population

| | | | TEATI | MENT GR | OUP (LT<br>N=XX | Γ2259 or V | isMed) | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Mild | | 1 | Modera | ite | | Sever | e |
| SOC and PT | ΑE | n | % | AE | n | % | ΑE | n | % |
| | (1) | (2) | (3) | (1) | (2) | (3) | (1) | (2) | (3) |
| Patients with at | | | | | | | | | |
| least one (*) | XX | xx | xx.x | XX | xx | xx.x | XX | xx | XX.X |
| SOC 1 | XX | xx | XX.X | XX | XX | XX.X | XX | xx | XX.X |
| SOC 1 – PT 1 | xx | xx | xx.x | xx | XX | xx.x | XX | XX | XX.X |
| SOC 1 – PT 2 | xx | XX | xx.x | XX | XX | xx.x | XX | XX | xx.x |
| | xx | XX | xx.x | XX | XX | XX.X | XX | xx | xx.x |

<sup>(1)</sup> Number of AEs: each AE is counted only once per SOC/PT

MedDRA version 22.0

SOC=System Organ Class, PT=Preferred Term, AE=Adverse Event.

Programming notes: replace (\*) by TEAE, ADE or SAD, depending on the table; when needed, update abbreviations;

Table xx: All TEAEs by SOC, PT and relationship (XX treatment group) – Safety population

| | TEATMENT GROUP (LT2259 or VisMed) | | | | | |
|---|---|---|---|---|---|---|
| | | | | N=XX | | |
| SOC and PT | Not | related t | o IMD | Re | lated to | IMD |
| | ΑE | n | % | AE | n | % |

<sup>(2)</sup> Number of subjects with at least one AE: each patient is counted only once per SOC/PT

<sup>(3) %</sup> of subjects with at least one AE

| | (1) | (2) | (3) | (1) | (2) | (3) |
|--------------|-----|-----|------|-----|-----|------|
| TOTAL | xx | XX | xx.x | xx | XX | xx.x |
| SOC 1 | xx | XX | xx.x | xx | XX | xx.x |
| SOC 1 – PT 1 | XX | XX | xx.x | xx | XX | XX.X |
| SOC 1 – PT 2 | XX | XX | xx.x | xx | XX | XX.X |
| | XX | XX | xx.x | xx | XX | XX.X |
| SOC 2 | XX | XX | xx.x | XX | XX | xx.x |
| SOC 2 – PT 1 | XX | XX | xx.x | XX | XX | XX.X |
| SOC 2 – PT 2 | XX | XX | xx.x | xx | XX | XX.X |
| •••• | XX | XX | xx.x | xx | XX | XX.X |

# 8 TABLES, LISTING AND FIGURES

#### 8.1 Planned tables

# Part 6.1 and 6.2: Disposition of patients

Table 1.1: First date and last date of selection visit, inclusion visit and last visit – All screened patients

Table 1.2: Number (%) of patients selected/not selected and reasons in case of non-selection – All screened patients

Table 1.3: Number (%) of patients who attended inclusion visit, number of patients included/not included and reasons in case of non-inclusion – Selected patients

Table 1.4: Number (%) of patients randomised/not randomised and reasons in case of non-randomisation – Included patients

Table 1.5: Number (%) of patients at each visit and type of last visit – Randomised patients

Table 1.6a: Number (%) of patients who completed the study and reasons in case of withdrawal – Randomised patients

Table 1.6b: Number (%) of patients who completed the study and reasons in case of withdrawal by possible impact of COVID-19 – SAF population

Table 1.6c: Number (%) of patients who completed the study and reasons in case of withdrawal by possible impact of COVID-19 – FAS population

Table 1.7a: Number (%) of patients in each population and reasons of exclusion – Randomised patients

Table 1.7b: Number (%) of patients in each population and reasons of exclusion by possible impact of COVID-19 – Randomised patients

Table 1.8a: Number (%) of patients in each country and site – FAS population

Table 1.8b: Number (%) of patients in each country and site by possible impact of COVID-19 – FAS population

Table 1.8c: Number (%) of patients in each country and site – SAF population

Table 1.8d: Number (%) of patients in each country and site by possible impact of COVID-19 – SAF population

Table 1.9: Time since inclusion for each visit – FAS population

Table 1.10: Study duration – FAS population

Table 1.11a: Protocol deviations – FAS population

Table 1.11b: Protocol deviations by possible impact of COVID-19 – FAS patient


### Part 6.3: Demographic and baseline characteristics

- Table 2.1a: Demographic characteristics PP population
- Table 2.1b: Demographic characteristics FAS population
- Table 2.1c: Demographic characteristics by possible impact of COVID-19 SAF population
- Table 2.1d: Demographic characteristics by possible impact of COVID-19 FAS population
- Table 2.2a: History of Dry Eye- PP population
- Table 2.2b: History of Dry Eye- FAS population
- Table 2.3a: Ocular medical history other than the studied disease by SOC and PT PP population
- Table 2.3b: Ocular medical history other than the studied disease by SOC and PT PP population
- Table 2.4a: Ocular medical surgery other than the studied disease by SOC and PT PP population
- Table 2.4b: Ocular medical surgery other than the studied disease by SOC and PT FAS populations
- Table 2.5a: Systemic medical history other than the studied disease by SOC and PT PP populations
- Table 2.5b: Systemic medical history other than the studied disease by SOC and PT FAS populations
- Table 2.6a: Systemic medical surgery other than the studied disease by SOC and PT PP population
- Table 2.6b: Systemic medical surgery other than the studied disease by SOC and PT FAS population

# Part 6.5: Previous and Concomitant Medications

- Table 3.1a: Previous ocular treatments by ATC level 2 and 4 PP population
- Table 3.1b: Previous ocular treatments (by ATC level 2 and 4) FAS population
- Table 3.2a: Concomitant ocular treatments (by ATC level 2 and 4) PP population
- Table 3.2b: Concomitant ocular treatments (by ATC level 2 and 4) FAS population
- Table 3.3a: Previous non-ocular treatments (by ATC level 2 and 4) PP population
- Table 3.3b: Previous non-ocular treatments (by ATC level 2 and 4) FAS population
- Table 3.4a: Concomitant non-ocular treatments (by ATC level 2 and 4) PP population
- Table 3.4b: Concomitant non-ocular treatments (by ATC level 2 and 4) FAS population
- Table 3.5a: Post-study treatments (by ATC level 2 and 4) PP population
- Table 3.5b: Post-study treatments (by ATC level 2 and 4) FAS population

### Part 6.6: Treatment exposure during the run-in period and IMD

- Table 4.1a: Treatment with Hyderabak duration in run-in period Safety population
- Table 4.1b: Treatment with Hyderabak duration in run-in period PP population
- Table 4.1c: Treatment with Hyderabak duration in run-in period FAS population

Table 4.2a: Time between last instillation of Hydrabak and inclusion visit date – Safety population

Table 4.2b: Time between last instillation of Hydrabak and inclusion visit date – PP population

Table 4.2c: Time between last instillation of Hydrabak and inclusion visit date – FAS population

Table 4.3a: Respect of dosage for Hydrabak – Safety population

Table 4.3b: Respect of dosage for Hydrabak – PP population

Table 4.3c: Respect of dosage for Hydrabak – FAS population

Table 4.4a: Study treatment duration – Safety population

Table 4.4b: Study treatment duration – PP population

Table 4.4c: Study treatment duration – FAS population

Table 4.5a: Mean daily dose regimen – Safety population

Table 4.5b: Mean daily dose regimen – PP population

Table 4.5c: Mean daily dose regimen – FAS population

## Part 6.7: Performance analysis

# Primary performance endpoint:

Table 5.1a: Oxford total score at each timepoint and change from baseline – Worst eye – PP population

Table 5.1b: Oxford total score at each timepoint and change from baseline – Worst eye – FAS population

Table 5.1c: Oxford total score at each timepoint and change from baseline – Worst eye – with LOCF imputation — FAS population

Table 5.2a: Oxford grade by panel at each timepoint and change from baseline – Worst eye – PP population

Table 5.2b: Oxford grade by panel at each timepoint and change from baseline – Worst eye – FAS population

Table 5.2c: Oxford grade by panel at each timepoint and change from baseline – Worst eye – with LOCF imputation — FAS population

Table 5.3a: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – (with country and country by treatment interaction) – PP population

Table 5.3b: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – (with country and country by treatment interaction) – FAS population

Table 5.3c: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – (with country and country by treatment interaction) – with LOCF imputation — FAS population

Table 5.4a: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye — PP population

Table 5.4b: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – as observed – FAS population

Table 5.4c: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – with LOCF imputation — FAS population

Table 5.5a: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – by possible impact of COVID-19 pandemic – PP population

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

Table 5.5b: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – by possible impact of COVID-19 pandemic – FAS population

Table 5.5c: Results of ANCOVA analysis in change from baseline in Oxford total score at D35 – Worst eye – by possible impact of COVID-19 pandemic – with LOCF imputation — FAS population

Table 5.6a: Results of MMRM analysis in change from baseline in Oxford total score at D35 – Worst eye – PP population

Table 5.6b: Results of MMRM analysis in change from baseline in Oxford total score at D35 – Worst eye – FAS population

Table 5.6c: Results of MMRM analysis in change from baseline in Oxford total score at D35 – Worst eye – with LOCF imputation — FAS population

# Secondary performance endpoints:

Table 5.7a: Results of ANCOVA analysis in change from baseline in Oxford total score at D8 and D84 – Worst eye – PP population

Table 5.7b: Results of ANCOVA analysis in change from baseline in Oxford total score at D8 and D84 – Worst eye – FAS population

Table 5.8a: Oxford total score at each timepoint and change from baseline – Contralateral eye – PP population

Table 5.8b: Oxford total score at each timepoint and change from baseline – Contralateral eye – FAS population

Table 5.9a: Oxford grade by panel at each timepoint and change from baseline – Contralateral eye – PP population

Table 5.9b: Oxford grade by panel at each timepoint and change from baseline – Contralateral eye – FAS population

Table 5.10a: Results of ANCOVA analysis in change from baseline in Oxford total score at D8, D35 and D84 – Contralateral eye – PP population

Table 5.10b: Results of ANCOVA analysis in change from baseline in Oxford total score at D8, D35 and D84 – Contralateral eye – FAS population

Table 5.11a: Van Bijsterveld items at each timepoint – Worst eye – PP population

Table 5.11b: Van Bijsterveld items at each timepoint – Worst eye – FAS population

Table 5.12a: Van Bijsterveld total score at each timepoint and change from baseline – Worst eye – PP population

Table 5.12b: Van Bijsterveld total score at each timepoint and change from baseline – Worst eye – FAS population

Table 5.13a: Van Bijsterveld – Results of ANCOVA analysis in change from baseline in Van Bijsterveld total score at D8, D35 and D84 – Worst eye – PP population

Table 5.13b: Van Bijsterveld – Results of ANCOVA analysis in change from baseline in Van Bijsterveld total score at D8, D35 and D84 – Worst eye – FAS population

Table 5.14a: Van Bijsterveld items at each timepoint – Contralateral eye – PP population Table 5.14b: Van Bijsterveld items at each timepoint – Contralateral eye – FAS population

Table 5.15a: Van Bijsterveld total score at each timepoint and change from baseline – Contralateral eye – PP population

Table 5.15b: Van Bijsterveld total score at each timepoint and change from baseline – Contralateral eye – FAS population

Table 5.16a: Van Bijsterveld – Results of ANCOVA analysis in change from baseline in Van Bijsterveld total score at D8, D35 and D84 – Contralateral eye – PP population

Table 5.16b: Van Bijsterveld – Results of ANCOVA analysis in change from baseline in Van Bijsterveld total score D8, D35 and D84 – Contralateral eye – FAS population

Table 5.17a: DEQ-5 items at each timepoint – PP population

Table 5.17b: DEQ-5 items at each timepoint – FAS population

Table 5.18a: DEQ-5 total score at each timepoint and change from baseline – PP population

Table 5.18b: DEQ-5 total score at each timepoint and change from baseline – FAS population

Table 5.19a: DEQ-5 – Results of ANCOVA analysis in change from baseline in DEQ-5 total score at D35 and D84 – PP population

Table 5.19b: DEQ-5 – Results of ANCOVA analysis in change from baseline in DEQ-5 total score at D35 and D84 – FAS population

Table 5.20a: OSDI items at each timepoint – PP population Table 5.20b: OSDI items at each timepoint – FAS population

Table 5.21a: OSDI total score at each timepoint and change from baseline – PP population Table 5.21b: OSDI total score at each timepoint and change from baseline – FAS population

Table 2.22a: OSDI – Results of ANCOVA analysis in change from baseline in OSDI total score at D8, D35 and D84 – PP population

Table 5.22b: OSDI – Results of ANCOVA analysis in change from baseline in OSDI total score at D8, D35 and D84 – FAS population

Table 5.23a: OSDI total score in classes at each timepoint – PP population Table 5.23b: OSDI total score in classes at each timepoint – FAS population

Table 5.24a: Schirmer test results at each timepoint and change from baseline – Worst eye – PP population

Table 5.24b: Schirmer test results at each timepoint and change from baseline – Worst eye – FAS population

Table 5.25a: Schirmer test – Results of ANCOVA analysis in change from baseline in Schirmer test at D8, D35 and D84 – Worst eye – PP population

Table 5.25b: Schirmer test – Results of ANCOVA analysis in change from baseline in Schirmer test at D8, D35 and D84 – Worst eye – FAS population

Table 5.26a: Schirmer test results at each timepoint and change from baseline – Contralateral eye – PP population

Table 5.26b: Schirmer test results at each timepoint and change from baseline – Contralateral eye – FAS population

Table 5.27a: Schirmer test – Results of ANCOVA analysis in change from baseline in Schirmer test at D8, D35 and D84 – Contralateral eye – PP population

Table 5.27b: Schirmer test – Results of ANCOVA analysis in change from baseline in Schirmer test at D8, D35 and D84 – Contralateral eye – FAS population

Table 5.28a: Measurements of TBUT at each timepoint – Worst eye – PP population Table 5.28b: Measurements of TBUT at each timepoint – Worst eye – FAS population

Table 5.29a: Mean TBUT at each timepoint and change from baseline – Worst eye – PP population

Table 5.29b: Mean TBUT at each timepoint and change from baseline – Worst eye – FAS population

Table 5.30a: Mean TBUT – Results of ANCOVA analysis in change from baseline in TBUT at D8, D35 and D84 – Worst eye – PP population

Table 5.30b: Mean TBUT – Results of ANCOVA analysis in change from baseline in TBUT at D8, D35 and D84 – Worst eye – FAS population

Table 5.31a: Measurements of TBUT at each timepoint – Contralateral eye – PP population Table 5.31b: Measurements of TBUT at each timepoint – Contralateral eye – FAS population

Table 5.32a: Mean TBUT at each timepoint and change from baseline – Contralateral eye – PP population

Table 5.32b: Mean TBUT at each timepoint and change from baseline – Contralateral eye – FAS population

Table 5.33a: Mean TBUT – Results of ANCOVA analysis in change from baseline in mean TBUT at D8, D35 and D84 – Contralateral eye – PP population

Table 5.33b: Mean TBUT – Results of ANCOVA analysis in change from baseline in mean TBUT at D8, D35 and D84 – Contralateral eye – FAS population

Table 5.34a: Conjunctival hyperaemia at each timepoint – Worst eye – PP population Table 5.34b: Conjunctival hyperaemia at each timepoint – Worst eye – FAS population

Table 5.35a: Conjunctival hyperaemia at each time point – Contralateral eye – PP population Table 5.35b: Conjunctival hyperaemia at each time point – Contralateral eye – FAS population

Table 5.36a: Dry eye symptoms at each timepoint – PP population Table 5.36b: Dry eye symptoms at each timepoint – FAS population

Table 5.37a: Dry eye symptoms total score at each timepoint and change from baseline – PP population

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

Table 5.37b: Dry eye symptoms total score at each timepoint and change from baseline – FAS population

Table 5.38a: Dry eye symptoms – Results of ANCOVA analysis in change from baseline in dry eye symptoms total score at D8, D35 and D84 – PP population

Table 5.38b: Dry eye symptoms – Results of ANCOVA analysis in change from baseline in dry eye symptoms total score at D8, D35 and D84 – FAS population

Table 5.39a: Performance assessment by the investigator at each time point – PP population Table 5.39b: Performance assessment by the investigator at each time point – FAS population

Table 5.40a: Quantification (AUF) and percentage of HLA-DR at each timepoint – PP population

Table 5.40b: Quantification (AUF) and percentage of HLA-DR at each timepoint – FAS population

Table 5.41a: Quantification (AUF) and percentage of HLA-DR in patients with severe dry eye at D84 – PP population

Table 5.41b: Quantification (AUF) and percentage of HLA-DR in patients with severe dry eye at D84 – FAS population

# Part 6.8: Safety analysis

### Safety endpoints:

Table 6.1: Ocular unusual sensation UPON INSTILLATION at least one time during the study—Safety population

Table 6.2: Ocular unusual sensation UPON INSTILLATION at each timepoint – Safety population Table 6.3: Ocular unusual sensation UPON INSTILLATION total score at each timepoint – Safety population

Table 6.4a: Far BCVA (in logMAR) at each timepoint – Worst eye – Safety population Table 6.4b: Far BCVA (/10) at each timepoint – Worst eye – Safety population

Table 6.5a: Far BCVA (in logMAR) at each timepoint – Contralateral eye – Safety population Table 6.5b: Far BCVA (/10) at each timepoint – Contralateral eye – Safety population

Table 6.6a: Tolerance assessment by the investigator at each timepoint – Safety population Table 6.6b: Tolerance assessment by the patient at each timepoint – Safety population

# Adverse events:

Table 6.7: Overview of ocular TEAEs – Safety population

Table 6.8: Overview of systemic TEAEs – Safety population

Table 6.9: Ocular TEAEs by SOC and PT – Safety population

Table 6.10: Non-ocular TEAEs by SOC and PT – Safety population


Table 6.11: Ocular non-serious TEAEs by SOC and PT – Safety population

Table 6.12: Systemic non-serious TEAEs by SOC and PT – Safety population

Table 6.13: Ocular treatment related TEAEs by SOC and PT – Safety Population

Table 6.14: Systemic treatment related TEAEs by SOC and PT – Safety Population

Table 6.15: Serious ocular TEAEs by SOC and PT – Safety population

Table 6.16: Serious systemic TEAEs by SOC and PT – Safety population

Table 6.17: Ocular TEAEs leading to medical device withdrawal by SOC and PT – Safety population

Table 6.18: Systemic TEAEs leading to medical device withdrawal by SOC and PT – Safety population

Table 6.19a: Ocular TEAEs by SOC, PT and severity (LT2259) – Safety population

Table 6.19b: Ocular TEAEs by SOC, PT and severity (Vismed) – Safety population

Table 6.20a: Systemic TEAEs by SOC, PT and severity (LT2259) – Safety population

Table 6.20b: Systemic TEAEs by SOC, PT and severity (Vismed) – Safety population

Table 6.21a: Ocular TEAEs by SOC, PT and relationship with the investigational medical device (LT2259) – Safety population

Table 6.21b: Ocular TEAEs by SOC, PT and relationship with the investigational medical device (Vismed) – Safety population

Table 6.22a: Systemic TEAEs by SOC, PT and relationship with the investigational medical device (LT2259) – Safety population

Table 6.22b: Systemic TEAEs by SOC, PT and relationship with the investigational medical device (Vismed) – Safety population

## 8.2 Planned listings

Listings 3 and 4 will include PP and FAS populations (as variable) and listing 5 will include FAS population.

# Part 6.2:

Listing 1: Non-selected patients, non-included patients and early withdrawals – All screened patients

Listing 2: Protocol deviations – FAS population

## Part 6.3:

Listing 3: Other aetiology of Dry Eye – Safety population

### Part 6.5:

Listing 4: Previous and concomitant treatments – Safety population

### Part 6.6:

Listing 5: Daily dose regimen different from 2 to 4 instillations/day – Safety population

#### Part 6.7:

Listing 6: OSI score – FAS population


#### Part 6.8:

Listing 7: Listing of individual data of overall systemic TEAEs – Safety population
Listing 8: Listing of individual data of overall ocular TEAEs – Safety population
Listing 9: Listing of individual data of overall systemic SAEs – Safety population
Listing 10: Listing of individual data of overall ocular SAEs – Safety population
Listing 11: Listing of individual data of overall systemic SADEs – Safety population
Listing 12: Listing of individual data of overall ocular SADEs – Safety population
Listing 13: Listing of individual data of non-emergent systemic AEs – Enrolled population
Listing 14: Listing of individual data of non-emergent ocular AEs – Enrolled population
Listing 15: Listing of COVID-19 AEs – Enrolled population

# 8.3 Planned figures

Figure 1: Flowchart

| Statistical analysis plan | 01JUL2021 |
|---------------------------|---------------|
| E876 | SAP Final 1.2 |

# 9 REFERENCES

NA.

#### 10 APPENDICES

### 10.1 Appendix 1: Level of validation for analyses programming

This chapter documents the validation of the statistical analysis programs. The level of validation is defined with reference to the procedure "Programming of the statistical analysis". All the analyses and programs have a default validation level "Basic + NC". Analysis below have a CR validation level:

| Analyses | Validation<br>level | Programs |
|--------------------------------------------|---------------------|-----------|
| Randomisation (when unblinding) | CR | FICH |
| Populations | CR | FICH |
| Derived data | CR | FICH |
| Primary efficacy endpoint (section 7.6.1) | CR | ANA_PRINC |
| Ocular unusual sensation UPON INSTILLATION | CR | ANA_SAFE |
| Adverse events | CR | ANA_SAFE |

## Key:

Basic = Corresponds to the self-check of the programming by any person who is required to program, as well as the checking of derived variables (see self-check frame)

NC (non-critical) = The tables, listings and figures compiled in a single document shall be verified by one qualified person other than the program developer with the support of the CRF and SAP for the study.

CR (critical) = A double programming and a comparison of the results should be performed by one qualified person other than the program developer.